CLINICAL TRIAL: NCT00555321
Title: Evaluation of Belatacept as First Line Immunosuppression in De Novo Liver Transplant Recipients
Brief Title: Belatacept in Liver Transplant Recipients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IM103-045
Record Dates: First submitted 2007-11-07; First posted 2007-11-08 (Estimated); Results first posted 2012-10-18 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-09

CONDITIONS: Immunosuppression in Solid Organ Transplant
MeSH Terms: interventions — Tacrolimus; Basiliximab; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group 1: Basiliximab+Belatacept (MI) + MMF (Experimental)
  Interventions: Drug: Basiliximab; Drug: Belatacept More Intensive (MI); Drug: Mycophenolate Mofetil (MMF)
- Group 2: Belatacept (MI) + MMF (Experimental)
  Interventions: Drug: Belatacept More Intensive (MI); Drug: Mycophenolate Mofetil (MMF)
- Group 3: Belatacept Less Intensive (LI) + MMF (Experimental)
  Interventions: Drug: Belatacept Less Intensive (LI); Drug: Mycophenolate Mofetil (MMF)
- Group 4: Tacrolimus + MMF (Other): Other
  Interventions: Drug: Tacrolimus; Drug: Mycophenolate Mofetil (MMF)
- Group 5: Tacrolimus (Active Comparator)
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — Capsules, Oral, dosed to achieve 12 hour trough level of 6-12 ng/mL, twice daily, 52 weeks (Short Term [ST]), in accordance with local practice and the package insert, 4 years (Long-Term Extension [LTE])
  Arms: Group 4: Tacrolimus + MMF; Group 5: Tacrolimus
Drug: Basiliximab — Intravenous (IV), 20 mg, Day1 and Day 5
  Arms: Group 1: Basiliximab+Belatacept (MI) + MMF
Drug: Belatacept More Intensive (MI) — Intravenous (IV),
  10 mg/kg on Days 1, 3 and 5, and at Weeks 2, 4, 6, 8, 10, 12, 16, 20, and 24.
  After 6 months (24 weeks) 5 mg/kg, every 4 weeks, 52 weeks (Short term [ST]), 5 mg/kg, every 4 weeks, 4 years (Long-term extension [LTE])
  Arms: Group 1: Basiliximab+Belatacept (MI) + MMF; Group 2: Belatacept (MI) + MMF
Drug: Belatacept Less Intensive (LI) — Intravenous (IV),
  10 mg/kg on Days 1, 3 and 5, and at Weeks 2, 4, 8 and 12.
  After 3 months (12 weeks) 5 mg/kg, every 4 weeks, 52 weeks (Short term [ST]), 5 mg/kg, every 4 weeks, 4 years (Long-Term Extension(LTE)
  Arms: Group 3: Belatacept Less Intensive (LI) + MMF
Drug: Mycophenolate Mofetil (MMF) — Intravenous (IV)/Capsules, IV/Oral, 1-2g/day, 52 weeks (Short term [ST]), ≤ 1 g/day, 4 years (Long-term extension [LTE])
  Arms: Group 1: Basiliximab+Belatacept (MI) + MMF; Group 2: Belatacept (MI) + MMF; Group 3: Belatacept Less Intensive (LI) + MMF; Group 4: Tacrolimus + MMF

SUMMARY:
The purpose of this clinical research study is to evaluate the effects of belatacept, relative to tacrolimus, on the incidence of rejection, graft loss and death in subjects receiving a liver transplant

ELIGIBILITY:
Inclusion Criteria:

* First time recipient of deceased donor liver transplant
* Age 18-70
* Hepatitis C virus (HCV) positive recipients
* For Long-term extension study-Subjects who have completed one year of study treatment (through Week 52)

Target Disease Exclusions:

Donor Exclusions a) Living donors b) ABO-incompatible donor recipient pairs c) Donor age < 12 or > 65 years d) Non heart-beating donors e) Anticipated cold ischemia time > 14 hours f) Donor Disease i) Known Human immunodeficiency virus (HIV) infection ii) Hepatitis B virus (HBV) surface antigen-positive or polymerase chain reaction (PCR)-positive donor if HBV negative recipient iii) HCV antibody-positive or PCR positive donor if HCV negative recipient

Recipient Exclusions g) Subjects with a history of hypercoagulable state h) Subjects with fulminant hepatic failure i) Subjects receiving a split or reduced liver j) Subjects who are Epstein-Barr virus (EBV) negative

Medical History and Concurrent Diseases

1. Subjects who have received 2 or more consecutive weeks of dialysis 1 month prior to enrollment OR anticipated to have prolonged dialysis post-transplantation
2. Subjects with known intrinsic renal disease (e.g., a urine protein/ creatinine ratio > 150 mg/g or the presence of an abnormal number of red blood cells (RBCs) or granular casts in the urine) AND calculated GFR < 40 ml/min/1.73 m^2 body surface area (BSA) (abbreviated Modification of Diet in Renal Disease [MDRD]). Subjects must have a calculated GFR assessment within 1 month prior to enrollment.
3. Subjects with known HIV
4. Subjects with any prior or concurrent solid organ (e.g., heart, kidney, pancreas) or cell (e.g., islet, bone marrow) transplant or subjects deemed likely to have a second solid organ or cell transplant (e.g., islet, bone marrow) within the next 3 years.
5. Subjects with a history of cancer within the last 5 years

Allergies and Adverse Drug Reactions

a) Hypersensitivity to any medications that will be used in the protocol

Prohibited Treatments and/or Therapies

1. Subjects receiving immunosuppressive agent(s) (e.g., methotrexate, abatacept, infliximab, etanercept, chemotherapy, etc.) within the past 6 months for other indications such as an autoimmune disease
2. Subjects who received maintenance corticosteroids at a dose of > 5 mg/day of prednisone (or equivalent) for at least 7 consecutive days within the prior year for an underlying chronic inflammatory or autoimmune disease
3. Subjects who have used any investigational drug within 30 days prior to the Day 1 visit
4. Subjects previously treated with belatacept

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2008-01; Primary Completion 2010-03 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (42):
- United States (19):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Usc University Hospital, Los Angeles, California
  - University Of California San Francisco Medical Center, San Francisco, California
  - Mayo Clinic Transplant Department, Jacksonville, Florida
  - Lifelink Healthcare Institute, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern University Feinberg School Of Medicine, Chicago, Illinois
  - Tulane Center For Abdominal Transplant, New Orleans, Louisiana
  - Henry Ford Hospital, Detriot, Michigan
  - University Of Minnesota, Minneapolis, Minnesota
  - Washington University School Of Medicine, St Louis, Missouri
  - Nyu School Of Medicine, New York, New York
  - Westchester Medical Center, Valhalla, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Univ. Of Cin. Coll. Of Med., Cincinnati, Ohio
  - Integris-Baptist Medical Ctr., Oklahoma City, Oklahoma
  - Hospital Of The University Of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor University Medical Center, Dallas, Texas
  - Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin
- Local Institution, Ciudad de Buenos Aires, Buenos Aires, Argentina
- Local Institution, Vienna, Austria
- Brazil (3):
  - Local Institution, Curitiba, Paraná
  - Local Institution, Rio de Janeiro, Rio de Janeiro
  - Local Institution, Centro-Porto Alegre, Rio Grande do Sul
- Canada (2):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Toronto, Ontario
- France (6):
  - Local Institution, Clichy
  - Local Institution, Lyon
  - Local Institution, Montpellier
  - Local Institution, Paris
  - Local Institution, Toulouse
  - Local Institution, Villejuif
- Germany (5):
  - Local Institution, Berlin
  - Local Institution, Hamburg
  - Local Institution, Hanover
  - Local Institution, Heidelberg
  - Local Institution, Tübingen
- Italy (4):
  - Local Institution, Bergamo
  - Local Institution, Padua
  - Local Institution, Pisa
  - Local Institution, Roma
- Local Institution, Barcelona, Spain

REFERENCES:
- [Derived] Klintmalm GB, Feng S, Lake JR, Vargas HE, Wekerle T, Agnes S, Brown KA, Nashan B, Rostaing L, Meadows-Shropshire S, Agarwal M, Harler MB, Garcia-Valdecasas JC. Belatacept-based immunosuppression in de novo liver transplant recipients: 1-year experience from a phase II randomized study. Am J Transplant. 2014 Aug;14(8):1817-27. doi: 10.1111/ajt.12810. PMID 25041339

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Basiliximab+Belatacept (MI) + MMF: Basiliximab- Intravenous (IV), 20 mg, on Day 1 and Day 5; Belatacept More Intensive (MI)-IV, 10 mg/kg on Days 1, 3 and 5, and at Weeks 2, 4, 6, 8, 10, 12, 16, 20 and 24. After 6 months (24 weeks) 5 mg/kg, every 4 weeks, 52 weeks (Short term [ST]), and 5 mg/kg, every 4 weeks, 4 years (Long-term extension [LTE]); Mycophenolate Mofetil (MMF)-IV/Capsules, IV/Oral, 1-2g/Day, 52 weeks (ST), and ≤ 1 g/Day, 4 years (LTE)
- Group 2: Belatacept (MI) + MMF: Belatacept MI- IV, 10 mg/kg on Days 1, 3 and 5, and at Weeks 2, 4, 6, 8, 10, 12, 16, 20, and 24. After 6 months (24 weeks) 5 mg/kg, every 4 weeks, 52 weeks (ST), and 5 mg/kg, every 4 weeks, 4 years (LTE); MMF-IV/Capsules, IV/Oral, 1-2g/Day, 52 weeks (ST), and ≤ 1 g/Day, 4 years (LTE)
- Group 3: Belatacept (LI) + MMF: Belatacept Less Intensive (LI)- IV, 10 mg/kg on Days 1, 3 and 5, and at Weeks 2, 4, 8 and 12. After 3 months (12 weeks) 5 mg/kg, every 4 weeks, 52 weeks (ST]), 5 mg/kg, every 4 weeks, 4 years (LTE); MMF, Intravenous (IV)/Capsules, IV/Oral, 1-2g/Day, 52 weeks (ST), ≤ 1 g/Day, 4 years (LTE)
- Group 4: Tacrolimus + MMF: Tacrolimus, Capsules, Oral, 6-12 ng/mL trough level, twice daily, 52 weeks (ST), in accordance with local practice and the package insert, 4 years (LTE); MMF, IV/Capsules, IV/Oral, 1-2g/Day, 52 weeks (ST), and ≤ 1 g/Day, 4 years (LTE)
- Group 5: Tacrolimus: Tacrolimus, Capsules, Oral, 6-12 ng/mL trough level, twice daily, 52 weeks (ST), in accordance with local practice and the package insert, and 4 years (LTE)
Period: Treatment Phase up to 12-months
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Started | 52 | 51 | 50 | 53 | 54
Received Transplant and Treated | 50 | 48 | 49 | 53 | 50
Completed | 31 | 29 | 26 | 46 | 32
Not Completed | 21 | 22 | 24 | 7 | 22
Not completed — Adverse Event | 6 | 7 | 11 | 7 | 18
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0 | 0
Not completed — Death | 2 | 1 | 4 | 0 | 0
Not completed — Lack of Efficacy | 9 | 8 | 5 | 0 | 0
Not completed — Other Reason | 1 | 3 | 2 | 0 | 0
Not completed — Never treated | 2 | 3 | 1 | 0 | 4
Period: Long-term Extension Phase
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Started | 30 (1 participant did not enter LTE) | 27 (2 participants did not enter LTE) | 24 (2 participants did not enter LTE) | 38 (8 participants did not enter LTE) | 26 (6 participants did not enter LTE)
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 30 | 27 | 24 | 38 | 26
Not completed — Adverse Event | 2 | 5 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 2 | 3 | 2
Not completed — Administrative reason by sponsor | 23 | 21 | 18 | 31 | 23
Not completed — Death | 2 | 0 | 0 | 3 | 0
Not completed — Participant did not meet study criteria | 0 | 0 | 0 | 0 | 1
Not completed — Other Reason | 1 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus | Total
Number analyzed (Participants) | 50 | 48 | 49 | 53 | 50 | 250
Age, Customized [Number; unit: participants]
  18 to 45 years | 7 | 7 | 4 | 11 | 4 | 33
  46 to 65 years | 41 | 40 | 43 | 37 | 42 | 203
  Above 65 years | 2 | 1 | 2 | 5 | 4 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 18 | 7 | 8 | 58
  Male | 39 | 34 | 31 | 46 | 42 | 192
Race/Ethnicity, Customized [Number; unit: participants]
  White | 44 | 40 | 46 | 49 | 43 | 222
  Black / African American | 4 | 3 | 1 | 3 | 2 | 13
  American Indian / Alaska native | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 1 | 0 | 2 | 0 | 0 | 3
  Other | 1 | 4 | 0 | 1 | 5 | 11
Race/Ethnicity, Customized [Number; unit: participants] — Ethnicity data collected in compliance with the 2005 Food and Drug Administration (FDA) Guidance for Industry for subjects enrolled in the United States (US) only.
  participants
    Hispanic or Latino (US sites) | 5 | 7 | 3 | 3 | 4 | 22
    Not Hispanic or Latino (US sites) | 28 | 16 | 11 | 22 | 23 | 100
    Unknown (Non- US sites) | 17 | 25 | 35 | 28 | 23 | 128
Model for End-Stage Liver Disease (MELD) score [Median (Full Range); unit: units on a scale] — The Model for End-Stage Liver Disease (MELD) is a scoring system for assessing the severity of chronic liver disease. MELD uses the participant's values for serum bilirubin, serum creatinine, and the international normalized ratio (INR) for prothrombin time to predict survival. 100% mortality= 3 month mortality is ≥ 40; 83% mortality= 3 month mortality 30-39; 76% mortality= 3 month mortality 20-29; 27% mortality= 3 month mortality 10-19; 4% mortality= 3 month mortality <10.
  units on a scale | 22.0 (8.19) [6.0 to 40.0] | 22.0 (8.29) [8.0 to 42.0] | 22.0 (6.05) [7.0 to 31.0] | 24.0 (7.48) [9.0 to 40.0] | 22.0 (5.48) [9.0 to 40.0] | 22.0 [6.0 to 42.0]
Primary cause of End Stage Liver Disease (ESLD) [Number; unit: participants]
  Non-cholestatic cirrhosis | 38 | 33 | 33 | 39 | 41 | 184
  Cholestatic liver disease cirrhosis | 0 | 3 | 3 | 1 | 2 | 9
  Biliary atresia | 0 | 0 | 0 | 1 | 0 | 1
  Acute hepatic necrosis | 4 | 0 | 3 | 1 | 0 | 8
  Metabolic disease | 0 | 2 | 0 | 1 | 0 | 3
  Malignant neoplasms | 4 | 7 | 5 | 6 | 3 | 25
  Other | 4 | 3 | 5 | 4 | 4 | 20
United Network for Organ Sharing (UNOS) Status [Number; unit: participants] — Participant's status category is determined by a point system, using objective and subjective factors. Status 1: critical, sudden liver failure, or newly transplanted liver not functioning; Status 2A: with chronic liver disease and are in the hospital's critical care unit. Status 1 and 2A have a life expectancy of less than 7 days without a liver transplant; Status 2B: with chronic liver disease, but do not meet the criteria for Status 2A; Status 3: with chronic liver disease, under continuous medical care, but not hospitalized, not meet the criteria for Status 2B.
  participants
    Status 1 | 0 | 1 | 0 | 0 | 0 | 1
    Status 2A | 1 | 1 | 2 | 3 | 0 | 7
    Status 2B | 3 | 2 | 5 | 1 | 2 | 13
    Status 3 | 2 | 2 | 2 | 1 | 1 | 8
    Not available | 44 | 42 | 40 | 48 | 47 | 221
Participants on Anti-Hypertensive Medications [Number; unit: participants]
  No | 41 | 39 | 41 | 42 | 40 | 203
  Yes | 9 | 9 | 8 | 11 | 10 | 47
Participants on Lipid Lowering Medications [Number; unit: participants]
  No | 46 | 43 | 48 | 51 | 44 | 232
  Yes | 4 | 5 | 1 | 2 | 6 | 18
Participants on Anti-diabetic Medications [Number; unit: participants]
  No | 35 | 35 | 40 | 41 | 38 | 189
  Yes | 15 | 13 | 9 | 12 | 12 | 61

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced at Least One Episode of Acute Rejection (AR), Graft Loss, or Death by 6 Months Post-transplant
Description: Any AR that was clinically suspected and biopsy proven (by central pathologist) was included in this triple composite end point. All biopsies for suspected AR were assessed by a blinded central histopathologist using Banff grading schema. Graft loss was defined as impairment of liver function to such a degree that the participant died or underwent re-transplantation. For 95% (confidence interval) CI within each group, normal approximation is used if N>=5, otherwise exact method is used.
Time Frame: At 6 months posttransplant
Population: Intent-to-Treat (ITT) population: all randomized and transplanted participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 50 | 48 | 49 | 53 | 50
percentage of participants | 48.0 [34.2 to 61.8] | 41.7 [27.7 to 55.6] | 46.9 [33.0 to 60.9] | 15.1 [5.5 to 24.7] | 38.0 [24.5 to 51.5]
Statistical Analysis 1: Comparison: Group 1: Basiliximab+Belatacept (MI) + MMF vs Group 4: Tacrolimus + MMF; Test type: Superiority or Other; Mean Difference (Final Values) = 32.9, 95% CI 2-sided [16.1 to 49.8] — For 95% CI of difference, adjustment was made for randomization strata (HCV-Infection status at baseline) if N >= 5 in each treatment arm. Otherwise exact method ignoring stratification was used
Statistical Analysis 2: Comparison: Group 2: Belatacept (MI) + MMF vs Group 4: Tacrolimus + MMF; Test type: Superiority or Other; Mean Difference (Final Values) = 26.6, 95% CI 2-sided [9.6 to 43.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Group 3: Belatacept (LI) + MMF vs Group 4: Tacrolimus + MMF; Test type: Superiority or Other; Mean Difference (Final Values) = 31.8, 95% CI 2-sided [14.8 to 48.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Group 1: Basiliximab+Belatacept (MI) + MMF vs Group 5: Tacrolimus; Test type: Superiority or Other; Mean Difference (Final Values) = 10.0, 95% CI 2-sided [-8.7 to 29.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Group 2: Belatacept (MI) + MMF vs Group 5: Tacrolimus; Test type: Superiority or Other; Mean Difference (Final Values) = 3.7, 95% CI 2-sided [-15.3 to 23.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Group 3: Belatacept (LI) + MMF vs Group 5: Tacrolimus; Test type: Superiority or Other; Mean Difference (Final Values) = 8.9, 95% CI 2-sided [-9.8 to 28.4] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Percentage of Participants Surviving With Functional Graft: 12-month Treatment Phase
Description: For 95% CI within each group, normal approximation was used if N>=5. Otherwise exact method was used.
Time Frame: At 6 and 12 months
Population: ITT population: all randomized and transplanted participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 50 | 48 | 49 | 53 | 50
percentage of participants
  At 6 months | 90.0 [81.7 to 98.3] | 89.6 [80.9 to 98.2] | 77.6 [65.9 to 89.2] | 92.5 [85.3 to 99.6] | 90.0 [81.7 to 98.3]
  At 12 months | 90.0 [81.7 to 98.3] | 83.3 [72.8 to 93.9] | 67.3 [54.2 to 80.5] | 92.5 [85.3 to 99.6] | 88.0 [79.0 to 97.0]
Statistical Analysis 1: Comparison: Group 1: Basiliximab+Belatacept (MI) + MMF vs Group 4: Tacrolimus + MMF; Analysis at Month 6; Test type: Superiority or Other; Mean Difference (Final Values) = -2.5, 95% CI 2-sided [-12.9 to 8.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Group 2: Belatacept (MI) + MMF vs Group 4: Tacrolimus + MMF; Analysis at Month 6; Test type: Superiority or Other; Mean Difference (Final Values) = -2.9, 95% CI 2-sided [-13.6 to 8.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Group 3: Belatacept (LI) + MMF vs Group 4: Tacrolimus + MMF; Analysis at Month 6; Test type: Superiority or Other; Mean Difference (Final Values) = -14.9, 95% CI 2-sided [-23.8 to 1.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Group 1: Basiliximab+Belatacept (MI) + MMF vs Group 5: Tacrolimus; Analysis at Month 6; Test type: Superiority or Other; Mean Difference (Final Values) = 0 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Group 2: Belatacept (MI) + MMF vs Group 5: Tacrolimus; Analysis at Month 6; Test type: Superiority or Other; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-12.1 to 11.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Group 3: Belatacept (LI) + MMF vs Group 5: Tacrolimus; Analysis at Month 6; Test type: Superiority or Other; Mean Difference (Final Values) = -12.4, 95% CI 2-sided [-22.9 to 4.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Group 1: Basiliximab+Belatacept (MI) + MMF vs Group 4: Tacrolimus + MMF; Analysis at Month 12; Test type: Superiority or Other; Mean Difference (Final Values) = -2.5, 95% CI 2-sided [-12.9 to 8.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Group 2: Belatacept (MI) + MMF vs Group 4: Tacrolimus + MMF; Analysis at Month 12; Test type: Superiority or Other; Mean Difference (Final Values) = -9.1, 95% CI 2-sided [-18.1 to 5.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Group 3: Belatacept (LI) + MMF vs Group 4: Tacrolimus + MMF; Analysis at Month 12; Test type: Superiority or Other; Mean Difference (Final Values) = -25.1, 95% CI 2-sided [-38.9 to -9.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Group 1: Basiliximab+Belatacept (MI) + MMF vs Group 5: Tacrolimus; Analysis at Month 12; Test type: Superiority or Other; Mean Difference (Final Values) = 2.0, 95% CI 2-sided [-9.9 to 14.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Group 2: Belatacept (MI) + MMF vs Group 5: Tacrolimus; Analysis at Month 12; Test type: Superiority or Other; Mean Difference (Final Values) = -4.7, 95% CI 2-sided [-15.5 to 10.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Group 3: Belatacept (LI) + MMF vs Group 5: Tacrolimus; Analysis at Month 12; Test type: Superiority or Other; Mean Difference (Final Values) = -20.7, 95% CI 2-sided [-35.5 to -4.1] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Participants Surviving With Functional Graft by End of Study (Includes LTE Data)
Description: For 95% CI within each group, normal approximation was used if N>=5, otherwise exact method was used.
Time Frame: Day 1 (randomization) through database lock (20-June-2011)
Population: ITT-LTE population, all randomized and transplanted participants who entered long term extension.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 30 | 27 | 24 | 38 | 26
percentage of participants | 93.3 [84.4 to 100.0] | 85.2 [71.8 to 98.6] | 95.8 [87.8 to 100.0] | 92.1 [83.5 to 100.0] | 96.2 [88.8 to 100.0]
Statistical Analysis 1: Comparison: Group 1: Basiliximab+Belatacept (MI) + MMF vs Group 4: Tacrolimus + MMF; Test type: Superiority or Other; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [-14.5 to 15.3] — For 95% CI of difference, normal approximation was used if N>=5 in both arms. Otherwise exact method was used
Statistical Analysis 2: Comparison: Group 2: Belatacept (MI) + MMF vs Group 4: Tacrolimus + MMF; Test type: Superiority or Other; Mean Difference (Final Values) = -6.9, 95% CI 2-sided [-25.7 to 8.8] — For 95% CI of difference, normal approximation was used if N>=5 in both arms. Otherwise exact method was used
Statistical Analysis 3: Comparison: Group 3: Belatacept (LI) + MMF vs Group 4: Tacrolimus + MMF; Test type: Superiority or Other; Mean Difference (Final Values) = 3.7, 95% CI 2-sided [-13.2 to 17.5] — For 95% CI of difference, normal approximation was used if N>=5 in both arms. Otherwise exact method was used
Statistical Analysis 4: Comparison: Group 1: Basiliximab+Belatacept (MI) + MMF vs Group 5: Tacrolimus; Test type: Superiority or Other; Mean Difference (Final Values) = -2.8, 95% CI 2-sided [-18.1 to 13.1] — For 95% CI of difference, normal approximation was used if N>=5 in both arms. Otherwise exact method was used
Statistical Analysis 5: Comparison: Group 2: Belatacept (MI) + MMF vs Group 5: Tacrolimus; Test type: Superiority or Other; Mean Difference (Final Values) = -11.0, 95% CI 2-sided [-29.4 to 6.2] — For 95% CI of difference, normal approximation was used if N>=5 in both arms. Otherwise exact method was used
Statistical Analysis 6: Comparison: Group 3: Belatacept (LI) + MMF vs Group 5: Tacrolimus; Test type: Superiority or Other; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-16.9 to 15.3] — For 95% CI of difference, normal approximation was used if N>=5 in both arms. Otherwise exact method was used

4. Secondary Outcome: Percentage of Participants Who Experienced at Least One Episode of Acute Rejection, Graft Loss, or Death by 12 Months
Description: Any AR that was clinically suspected and biopsy proven (by central pathologist) was included in this triple composite end point. All biopsies for suspected AR were assessed by a blinded central histopathologist using Banff grading. Graft loss was defined as impairment of liver function to such a degree that the participant died or underwent re-transplantation. For 95% CI within each group, normal approximation is used if N>=5. Otherwise exact method is used. For 95% CI of difference, adjustment is made for randomization strata if N >= 5 in each treatment arm.
Time Frame: At 12 months posttransplant
Population: ITT population: all randomized and transplanted participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 50 | 48 | 49 | 53 | 50
percentage of participants | 52.0 [38.2 to 65.8] | 47.9 [33.8 to 62.0] | 53.1 [39.1 to 67.0] | 18.9 [8.3 to 29.4] | 40.0 [26.4 to 53.6]
Statistical Analysis 1: Comparison: Group 1: Basiliximab+Belatacept (MI) + MMF vs Group 4: Tacrolimus + MMF; Test type: Superiority or Other; Mean Difference (Final Values) = 33.1, 95% CI 2-sided [15.8 to 50.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Group 2: Belatacept (MI) + MMF vs Group 4: Tacrolimus + MMF; Test type: Superiority or Other; Mean Difference (Final Values) = 29.0, 95% CI 2-sided [11.4 to 46.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Group 3: Belatacept (LI) + MMF vs Group 4: Tacrolimus + MMF; Test type: Superiority or Other; Mean Difference (Final Values) = 34.2, 95% CI 2-sided [16.9 to 51.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Group 1: Basiliximab+Belatacept (MI) + MMF vs Group 5: Tacrolimus; Test type: Superiority or Other; Mean Difference (Final Values) = 12.0, 95% CI 2-sided [-7.1 to 31.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Group 2: Belatacept (MI) + MMF vs Group 5: Tacrolimus; Test type: Superiority or Other; Mean Difference (Final Values) = 7.9, 95% CI 2-sided [-11.5 to 27.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Group 3: Belatacept (LI) + MMF vs Group 5: Tacrolimus; Test type: Superiority or Other; Mean Difference (Final Values) = 13.1, 95% CI 2-sided [-5.9 to 32.6] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Percentage of Participants Who Experienced at Least One Episode of Acute Rejection, Graft Loss, or Death by End of Study (Includes LTE Data)
Description: Any AR that was clinically suspected and biopsy proven (by central pathologist) was included in this triple composite end point. All biopsies for suspected AR were assessed by a central histopathologist using Banff criteria. For 95% CI within each group, normal approximation was used if N>=5, otherwise exact method was used.
Time Frame: Day 1 (randomization) through database lock (20-June-2011)
Population: ITT-LTE population: all randomized and transplanted participants who entered the Long term extension
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 30 | 27 | 24 | 38 | 26
percentage of participants | 36.7 [19.4 to 53.9] | 37.0 [18.8 to 55.3] | 25.0 [7.7 to 42.3] | 21.1 [8.1 to 34.0] | 23.1 [6.9 to 39.3]
Statistical Analysis 1: Comparison: Group 1: Basiliximab+Belatacept (MI) + MMF vs Group 4: Tacrolimus + MMF; Test type: Superiority or Other; Mean Difference (Final Values) = 15.6, 95% CI 2-sided [-5.8 to 36.8] — For 95% CI of difference, normal approximation was used if N>=5 in both arms. Otherwise exact method was used
Statistical Analysis 2: Comparison: Group 2: Belatacept (MI) + MMF vs Group 4: Tacrolimus + MMF; Test type: Superiority or Other; Mean Difference (Final Values) = 16.0, 95% CI 2-sided [-6.0 to 38.0] — For 95% CI of difference, normal approximation was used if N>=5 in both arms. Otherwise exact method was used
Statistical Analysis 3: Comparison: Group 3: Belatacept (LI) + MMF vs Group 4: Tacrolimus + MMF; Test type: Superiority or Other; Mean Difference (Final Values) = 3.9, 95% CI 2-sided [-16.6 to 26.8] — For 95% CI of difference, normal approximation was used if N>=5 in both arms. Otherwise exact method was used
Statistical Analysis 4: Comparison: Group 1: Basiliximab+Belatacept (MI) + MMF vs Group 5: Tacrolimus; Test type: Superiority or Other; Mean Difference (Final Values) = 13.6, 95% CI 2-sided [-10.8 to 36.1] — For 95% CI of difference, normal approximation was used if N>=5 in both arms. Otherwise exact method was used
Statistical Analysis 5: Comparison: Group 2: Belatacept (MI) + MMF vs Group 5: Tacrolimus; Test type: Superiority or Other; Mean Difference (Final Values) = 14.0, 95% CI 2-sided [-10.9 to 37.3] — For 95% CI of difference, normal approximation was used if N>=5 in both arms. Otherwise exact method was used
Statistical Analysis 6: Comparison: Group 3: Belatacept (LI) + MMF vs Group 5: Tacrolimus; Test type: Superiority or Other; Mean Difference (Final Values) = 1.9, 95% CI 2-sided [-21.8 to 26.0] — For 95% CI of difference, normal approximation was used if N>=5 in both arms. Otherwise exact method was used

6. Secondary Outcome: Number of Participants Having Acute Rejections: 12-month Treatment Phase
Description: Acute rejections were clinically suspected and biopsy proven by central pathologist. The number of episodes of AR was counted.
Time Frame: 3 , 6, and 12 months
Population: ITT population: all randomized and transplanted participants
Measure: Number; unit: participants
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 50 | 48 | 49 | 53 | 50
participants
  By 3 months ; Overall | 17 | 15 | 14 | 4 | 13
  By 3 months ; 1 episode | 15 | 14 | 14 | 4 | 12
  By 3 months ; 2 episodes | 1 | 1 | 0 | 0 | 1
  By 3 months ; >2 episodes | 1 | 0 | 0 | 0 | 0
  By 6 months ; Overall | 20 | 15 | 15 | 5 | 15
  By 6 months ; 1 episode | 18 | 12 | 14 | 4 | 13
  By 6 months ; 2 episodes | 1 | 3 | 1 | 1 | 2
  By 6 months ; >2 episodes | 1 | 0 | 0 | 0 | 0
  By 12 months ; Overall | 22 | 16 | 16 | 7 | 15
  By 12 months ; 1 episode | 18 | 13 | 14 | 6 | 13
  By 12 months ; 2 episodes | 3 | 3 | 2 | 1 | 2
  By 12 months ; >2 episodes | 1 | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants Having Acute Rejections During the LTE
Description: as for outcome 6
Time Frame: Day 1 (randomization) through database lock (20-June-2011)
Population: ITT-LTE population, all randomized and transplanted participants who entered long-term extension
Measure: Number; unit: participants
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 30 | 27 | 24 | 38 | 26
participants
  By 12 months (m); Overall | 9 | 6 | 6 | 6 | 6
  By 12 m ; 1 episode | 8 | 6 | 5 | 5 | 5
  By 12 m ; 2 episodes | 1 | 0 | 1 | 1 | 1
  By 12 m; >2 episodes | 0 | 0 | 0 | 0 | 0
  By Database lock; Overall | 9 | 6 | 6 | 6 | 6
  By Database lock ; 1 episode | 8 | 6 | 5 | 5 | 5
  By Database lock ; 2 episodes | 1 | 0 | 1 | 1 | 0
  By Database lock ; >2 episodes | 0 | 0 | 0 | 0 | 1

8. Secondary Outcome: Number of Participants With Central Biopsy Proven Acute Rejection by Treatment Type by 12 Months
Description: Acute rejections were clinically suspected and biopsy proven by central pathologist. Corticosteroid-resistant rejection = Continued rejection, as documented by liver biopsy, after the completion of 2 days of corticosteroids and requiring use of T-cell depleting agent. Refractory rejection=Continued rejection, as documented by liver biopsy, after use of corticosteroids and T cell depletion therapy. Increase in the dose of TAC was monitored in participants who were assigned to one of the TAC-based regimens. TRT= treatment
Time Frame: 3, 6 and 12 months posttransplant
Population: ITT population: all randomized and transplanted participants
Measure: Number; unit: participants
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 50 | 48 | 49 | 53 | 50
participants
  By 3 months: Acute rejections | 7 | 15 | 14 | 4 | 13
  By 3 months: Treated participants | 10 | 11 | 7 | 3 | 10
  By 3 months: Corticosteroid treatment Only | 10 | 7 | 7 | 2 | 9
  By 3 months: Corticosteroid resistant | 0 | 1 | 0 | 0 | 0
  By 3 months: Refractory | 0 | 1 | 0 | 0 | 0
  By3 months: Initial lymphocyte depleting TRT | 0 | 2 | 0 | 0 | 0
  By 3 months: Increase in dose of Tacrolimus | 0 | 0 | 0 | 1 | 1
  By 3 months: Other / not available | 0 | 0 | 0 | 0 | 0
  By 6 months: Acute rejections | 20 | 15 | 15 | 5 | 15
  By 6 months: Treated participants | 12 | 11 | 8 | 4 | 12
  By 6 months: Corticosteroid treatment Only | 12 | 6 | 8 | 3 | 10
  By 6 months: Corticosteroid resistant | 0 | 1 | 0 | 0 | 0
  By 6 months: Refractory | 0 | 1 | 0 | 0 | 0
  By 6 months: Initial lymphocyte depleting TRT | 0 | 3 | 0 | 0 | 0
  By 6 months: Increase in dose of Tacrolimus | 0 | 0 | 0 | 1 | 1
  By 6 months: Other / not available | 0 | 0 | 0 | 0 | 1
  By 12 months: Acute rejections | 22 | 16 | 16 | 7 | 15
  By 12 months: Treated participants | 12 | 12 | 8 | 5 | 2
  By 12 months: Corticosteroid treatment Only | 12 | 7 | 8 | 4 | 10
  By 12 months: Corticosteroid resistant | 0 | 1 | 0 | 0 | 0
  By 12 months: Refractory | 0 | 1 | 0 | 0 | 0
  B12 months: Initial lymphocyte depleting TRT | 0 | 3 | 0 | 0 | 0
  12 months: Other / not available | 0 | 0 | 0 | 0 | 1

9. Secondary Outcome: Number of Participants With Central Biopsy Proven Acute Rejection by Treatment Type During the LTE
Description: Acute rejections were clinically suspected and biopsy proven by central pathologist. Corticosteroid-resistant rejection = Continued rejection, as documented by liver biopsy, after the completion of 2 days of corticosteroids and requiring use of T-cell depleting agent. Refractory rejection=Continued rejection, as documented by liver biopsy, after use of corticosteroids and T cell depletion therapy. Increase in the dose of TAC was monitored in participants who were assigned to one of the TAC-based regimens. DBL=database lock, TRT=treatment
Time Frame: Day 1 (randomization) through database lock (20-June-2011)
Population: ITT-LTE population, all randomized and transplanted participants who entered long term extension.
Measure: Number; unit: participants
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 30 | 27 | 24 | 38 | 26
participants
  By 12 months: Acute rejections | 9 | 6 | 6 | 6 | 6
  By 12 months: Treated participants | 4 | 5 | 4 | 5 | 6
  By 12 months: Corticosteroid treatment Only | 4 | 4 | 4 | 4 | 5
  By 12 months: Corticosteroid resistant | 0 | 0 | 0 | 0 | 0
  By 12 months: Refractory | 0 | 0 | 0 | 0 | 0
  By 12 months: Initial lymphocyte depleting TRT | 0 | 1 | 0 | 0 | 0
  By 12 months: Other / not available | 0 | 0 | 0 | 0 | 0
  By 12 months: Increase in dose of TAC | 0 | 0 | 0 | 1 | 0
  By DBL: Acute rejections | 9 | 6 | 6 | 6 | 6
  By DBL: Treated participants | 4 | 5 | 4 | 5 | 6
  By DBL: Corticosteroid treatment Only | 4 | 4 | 4 | 4 | 5
  By DBL: Corticosteroid resistant | 0 | 0 | 0 | 0 | 0
  By DBL: Refractory | 0 | 0 | 0 | 0 | 0
  By DBL: Initial lymphocyte depleting treatment | 0 | 1 | 0 | 0 | 0
  By DBL: Other/ Not available | 0 | 0 | 0 | 0 | 0
  By DBL: Increase in dose of TAC | 0 | 0 | 0 | 1 | 1

10. Secondary Outcome: Number of Participants Who Had Acute Rejection by Banff Grade by 12 Months
Description: Acute Rejections (AR) were clinically suspected and biopsy proven by central pathologist. The Banff grading is a classification of renal allograft pathology and AR. Grade I: AR requiring moderate (>25%) to severe mononuclear cell interstitial infiltrate and moderate tubulitis; Grade II: AR requiring severe tubulitis and/or intimal arteritis; Grade III: AR requiring transmural arteritis. Only the episode with highest Banff grade for each participant was counted.
Time Frame: 3, 6 and 12 months posttransplant
Population: ITT population: all randomized and transplanted participants
Measure: Number; unit: participants
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 50 | 48 | 49 | 53 | 50
participants
  By 3 months: Grade 1 | 14 [20.9 to 47.1] | 8 [18.1 to 44.4] | 7 [15.9 to 41.2] | 3 [2.1 to 18.2] | 6 [13.8 to 38.2]
  By 3 months: Grade 2 | 3 [26.4 to 53.6] | 6 [18.1 to 44.4] | 6 [17.7 to 43.5] | 1 [1.6 to 17.3] | 5 [17.3 to 42.7]
  By 3 months: Grade 3 | 0 [30.2 to 57.8] | 1 [20.0 to 46.7] | 1 [19.5 to 45.8] | 0 [4.1 to 22.3] | 2 [17.3 to 42.7]
  By 6 months: Grade 1 | 16 | 6 | 7 | 4 | 7
  By 6 months: Grade 2 | 4 | 8 | 7 | 1 | 6
  By 6 months: Grade 3 | 0 | 1 | 1 | 0 | 2
  By 12 months: Grade 1 | 15 | 7 | 7 | 6 | 7
  By 12 months: Grade 2 | 7 | 8 | 8 | 1 | 6
  By 12 months: Grade 3 | 0 | 1 | 1 | 0 | 2

11. Secondary Outcome: Number of Participants With Acute Rejections by Rejection Activity Index (RAI) by 12 Months
Description: Acute Rejections were clinically suspected and biopsy proven by central pathologist. The Banff Rejection Activity Index (RAI) comprises 3 components scored from 0 to 3: venous endothelial inflammation; bile duct inflammation damage; and portal inflammation; the scores are combined to an overall score (the RAI). An overall score of 0-2 is considered indeterminate, score of 3-4 is mild, score of 5-6 is moderate, and score of 7-9 is severe. Only the episode with the highest total RAI score for each participant was counted.
Time Frame: 3, 6 and 12 months posttransplant
Population: ITT population: all randomized and transplanted participants
Measure: Number; unit: participants
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 50 | 48 | 49 | 53 | 50
participants
  By 3 months; Indeterminate score | 0 | 0 | 0 | 0 | 0
  By 3 months; Mild Score | 14 | 8 | 7 | 3 | 7
  By 3 months; Moderate Score | 3 | 6 | 7 | 1 | 2
  By 3 months; Severe Score | 0 | 1 | 0 | 0 | 4
  By 6 months; Indeterminate score | 0 | 0 | 0 | 0 | 0
  By 6 months; Mild Score | 17 | 6 | 7 | 4 | 8
  By 6 months; Moderate Score | 3 | 8 | 8 | 1 | 3
  By 6 months; Severe Score | 0 | 1 | 0 | 0 | 4
  By 12 months; Indeterminate score | 0 | 0 | 0 | 0 | 0
  By 12 months; Mild Score | 17 | 7 | 7 | 6 | 8
  By 12 months; Moderate Score | 4 | 8 | 9 | 1 | 3
  By 12 months; Severe Score | 1 | 1 | 0 | 0 | 4

12. Secondary Outcome: Number of Participants Having Acute Rejection by Rejection Activity Index During the LTE
Description: as for outcome 11
Time Frame: Day 1 (randomization) through End of study (database lock of 20-June-2011)
Population: ITT-LTE population, all randomized and transplanted participants who entered the long-term extension phase.
Measure: Number; unit: participants
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 30 | 27 | 24 | 38 | 26
participants
  By 12 months; Indeterminate score | 0 | 0 | 0 | 0 | 0
  By 12 months; Mild Score | 8 | 5 | 2 | 5 | 4
  By 12 months; Moderate Score | 1 | 1 | 4 | 1 | 0
  By 12 months; Severe Score | 0 | 0 | 0 | 0 | 2
  At end of study; Indeterminate score | 0 | 0 | 0 | 0 | 0
  At end of study; Mild Score | 8 | 5 | 2 | 5 | 4
  At end of study; Moderate Score | 1 | 1 | 4 | 1 | 0
  At end of study; Severe Score | 0 | 0 | 0 | 0 | 2

13. Secondary Outcome: Number of Participants at Risk of First Acute Rejection as Determined by Kaplan-Meier Method by 12 Months
Description: The time from transplantation to the first AR episode in each treatment arm was summarized using Kaplan-Meier curves. Acute Rejections were clinically suspected and biopsy proven by central pathologist.
Time Frame: 3, 6, 9 and 12 months posttransplant
Population: ITT population, all randomized and transplanted participants.
Measure: Number; unit: participants
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 50 | 48 | 49 | 53 | 50
participants
  By 3 months | 30 | 31 | 30 | 48 | 34
  By 6 months | 27 | 29 | 28 | 47 | 32
  By 9 months | 25 | 29 | 27 | 47 | 32
  By 12 months | 23 | 25 | 23 | 42 | 28

14. Secondary Outcome: Mean Change From Baseline in Measured Glomerular Filtration Rate (GFR): 12-month Treatment Phase
Description: GFR was assessed using a true measure of glomerular filtration via iothalamate clearance test. The month 2 time point was selected as the "baseline" time point with respect to measured GFR due to logistical difficulty in obtaining measured GFR at the time of liver transplant and post-transplant renal function largely stabilizing by 2 months. All Measured GFR > 200 were truncated at 200.
Time Frame: Baseline (2 month), 12 months posttransplant
Population: ITT population: all randomized and transplanted subjects. n = participants who had both baseline and postbaseline values.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 50 | 48 | 49 | 53 | 50
mL/min/1.73m^2
  2 months (n=37, 36, 35, 41, 37) | 72.4 (29.50) | 86.6 (37.38) | 98.6 (41.89) | 65.9 (35.52) | 58.5 (33.96)
  12 months (n=39, 35, 29, 40, 32) | 88.9 (36.34) | 93.1 (38.99) | 73.1 (36.82) | 75.2 (46.89) | 70.5 (29.59)
  Change from 2 to 12 months (n=31, 29, 26, 36, 29) | 14.2 (40.64) | 5.8 (48.20) | -19.6 (49.56) | 5.3 (51.81) | 7.3 (31.59)

15. Secondary Outcome: Mean Change From Baseline in Calculated GFR, by Modification of Diet in Renal Disease (MDRD) Equation: 12-month Treatment Phase
Description: GFR is a measure of the rate at which blood is filtered by the kidney. MDRD is an equation (calculation) used to estimate GFR in participants with impaired renal function based on serum creatinine (ScR), age, race, gender, blood urea nitrogen (BUN), and albumin (Alb). GFR (mL/min/1.73 m^2) = 170*(Scr)^-0.999*(Age)^-0.176*(0.762 if female)*(1.180 if African American)*(BUN)^-0.170*(Alb)^+0.318. ). BL= baseline, mL= milliliters; min= minute; m^2= meters squared.
Time Frame: Baseline [BL] (pretransplant time point), 1, 2, 3, 6 and 12 months posttransplant
Population: ITT population, all randomized and transplanted participants. n = participants who had both baseline and postbaseline values.
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 50 | 48 | 49 | 53 | 50
mL/min/1.73 m^2
  BL; (n=47, 42, 42, 45, 45) | 66.3 (29.14) | 77.4 (33.42) | 76.6 (27.77) | 73.7 (32.42) | 80.2 (30.78)
  1 month; (n=45, 44, 42, 49, 49) | 85.6 (25.27) | 93.1 (35.66) | 89.6 (28.47) | 64.9 (26.31) | 62.2 (31.94)
  Change from BL to 1 month; (n=43, 38, 37, 41, 45) | 21.0 (33.76) | 15.3 (44.72) | 11.4 (31.34) | -8.7 (33.91) | -17.7 (40.65)
  2 months; (n=29, 30, 23, 25, 27) | 86.1 (21.78) | 96.6 (27.78) | 105.8 (31.98) | 76.3 (35.25) | 66.9 (28.42)
  Change from BL to 2 months; (n=28, 26, 20, 22, 25) | 25.3 (32.35) | 18.3 (33.35) | 31.5 (26.89) | -1.5 (52.78) | -14.0 (34.03)
  3 months; (n=36, 36, 35, 46, 37) | 86.5 (21.20) | 91.7 (26.83) | 96.6 (27.02) | 65.0 (19.93) | 60.4 (22.98)
  Change from BL to 3 months; (n=33, 34, 30, 40, 33) | 22.0 (29.04) | 13.3 (31.50) | 18.3 (26.92) | -8.4 (30.89) | -20.2 (32.08)
  6 months; (n=39, 34, 38, 49, 36) | 82.2 (23.88) | 90.3 (24.23) | 86.0 (28.74) | 61.9 (20.62) | 59.8 (22.37)
  Change from BL to 6 months; (n=37, 30, 33, 42, 31) | 18.6 (31.06) | 7.6 (31.43) | 5.6 (26.78) | -11.7 (30.61) | -22.7 (29.63)
  12 months; (n=40, 33, 35, 46, 38) | 83.8 (22.18) | 97.7 (23.80) | 85.6 (31.23) | 68.4 (26.09) | 63.8 (21.24)
  Change from BL to 12 month; (n=37, 29, 30, 41, 33) | 18.2 (27.63) | 19.2 (30.05) | 4.2 (30.40) | -6.3 (40.08) | -17.1 (28.61)

16. Secondary Outcome: Mean Change From Baseline in Calculated GFR During the LTE
Description: as for outcome 15
Time Frame: Baseline (pretransplant time point), 1, 2, 3, 6,12, 18, 24, 30, 36 months posttransplant
Population: ITT-LTE population, all randomized and transplanted participants who entered long term extension. n= participants who have both baseline and postbaseline values.
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 30 | 27 | 24 | 38 | 26
mL/min/1.73 m^2
  Baseline (BL); (n=27,24,20,33,23) | 64.4 (32.98) | 85.6 (34.74) | 78.0 (31.65) | 77.9 (32.13) | 83.0 (35.80)
  1 month; (n=28,27,23,36,25) | 88.2 (24.56) | 103.1 (38.89) | 95.1 (26.70) | 68.6 (28.06) | 59.1 (22.41)
  Change from BL to 1 month; (n=26,24,20,31,23) | 26.3 (30.52) | 20.2 (52.60) | 16.0 (31.53) | -7.6 (37.19) | -22.6 (25.62)
  2 months; (n=21,21,15,19,19) | 86.2 (22.29) | 99.4 (29.58) | 102.3 (32.44) | 71.2 (18.88) | 64.4 (28.90)
  Change from BL to 2 months; (n=20,19,14,17,18) | 26.0 (34.74) | 12.6 (30.12) | 30.7 (29.13) | -11.6 (36.28) | -17.4 (33.94)
  3 months; (n=27, 26, 24, 35, 24) | 87.0 (22.30) | 97.0 (26.14) | 97.0 (25.94) | 66.5 (20.36) | 57.0 (22.61)
  Change from BL to 3 months; (n=24, 24, 20, 30, 21) | 23.3 (32.20) | 13.7 (32.38) | 17.0 (27.99) | -8.1 (31.69) | -23.5 (30.57)
  6 months; (n=29, 26, 24, 24, 38, 23) | 87.6 (23.93) | 93.1 (23.45) | 92.3 (24.71) | 64.6 (20.43) | 56.7 (20.37)
  Change from BL to 6 months; (n=27, 23, 20, 33, 20) | 24.0 (33.34) | 8.6 (31.89) | 12.2 (21.59) | -10.9 (30.53) | -23.3 (28.74)
  12 months; (n=29, 25, 24, 36, 24) | 88.1 (21.45) | 101.3 (25.01) | 94.8 (27.89) | 67.8 (22.07) | 61.7 (20.49)
  Change from BL to 12 months; (n=26, 23, 20, 31,21) | 22.6 (29.57) | 19.4 (30.28) | 16.5 (24.91) | -9.3 (34.30) | -20.2 (27.65)
  18 months; (n=24, 25, 21, 33, 21) | 84.8 (24.10) | 95.0 (24.54) | 91.3 (25.35) | 69.0 (22.84) | 63.2 (21.25)
  Change from BL to 18 months; (n=21, 23, 17, 28,18) | 22.5 (34.16) | 11.2 (34.07) | 7.4 (20.11) | -6.8 (31.26) | -6.1 (22.80)
  24 months; (n=13, 15, 15, 22, 15) | 84.8 (26.18) | 87.6 (21.43) | 96.3 (26.02) | 73.3 (22.82) | 66.3 (21.63)
  Change from BL to 24 months; (n=10, 13, 11, 19,13) | 27.9 (33.76) | 9.9 (37.62) | 15.2 (19.64) | -2.2 (32.67) | 2.3 (24.58)
  At 30 months; (n=6, 6, 6, 12, 7) | 102.9 (20.92) | 94.4 (31.78) | 90.4 (22.76) | 64.1 (27.30) | 59.5 (20.47)
  Change from BL to 30 months; (n=5, 5, 3, 8, 6) | 41.4 (33.98) | 40.4 (38.10) | 17.1 (26.76) | -15.0 (38.89) | -10.7 (13.40)

17. Secondary Outcome: Mean Change From Baseline Serum Creatinine at Months 1, 2, 3, 6 and 12
Description: Measurement of SCr is commonly used as an indicator of renal function. High creatinine blood level is an indicator of deficient filtering by the kidney. SCr was determined at baseline and various post-baseline time points.
Time Frame: Baseline (pretransplant time point), 1, 2, 3, 6 and 12 months posttransplant
Population: ITT population, all randomized and transplanted participants. n= participants who have both baseline and postbaseline values.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 50 | 48 | 49 | 53 | 50
mg/dL
  Baseline (BL); (n=47, 42, 42, 45, 45) | 1.4 (1.25) | 1.0 (0.39) | 0.9 (0.38) | 1.1 (0.54) | 1.0 (0.40)
  At 1 months; (n=45, 44, 42, 49, 49) | 0.9 (0.38) | 0.8 (0.32) | 0.9 (0.42) | 1.2 (0.41) | 1.3 (0.68)
  Change from BL to 1 months; (n=43, 38, 37, 41, 45) | -0.5 (1.35) | -0.1 (0.50) | -0.1 (0.48) | 0.1 (0.52) | 0.3 (0.75)
  At 2 months; (n=29, 30, 23, 25, 27) | 0.9 (0.21) | 0.8 (0.22) | 0.8 (0.28) | 1.0 (0.30) | 1.2 (0.36)
  Change from BL to 2 months; (n=28, 26, 20, 22, 25) | -0.7 (1.54) | -0.2 (0.32) | -0.2 (0.32) | 0.0 (0.73) | 0.2 (0.45)
  At 3 months; (n=36, 36, 35, 46, 37) | 0.9 (0.27) | 0.9 (0.21) | 0.8 (0.24) | 1.2 (0.36) | 1.3 (0.53)
  Change from BL to 3 months; (n=33, 34, 30, 40, 33) | -0.6 (1.45) | -0.1 (0.44) | -0.1 (0.32) | 0.1 (0.50) | 0.3 (0.42)
  At 6 months; (n=39, 34, 38, 49, 36) | 1.0 (0.30) | 0.9 (0.20) | 0.9 (0.42) | 1.3 (0.44) | 1.3 (0.51)
  Change from BL to 6 months; (n=37, 30, 33, 42, 31) | -0.5 (1.39) | 0.0 (0.41) | 0.1 (0.43) | 0.2 (0.60) | 0.4 (0.50)
  At 12 months; (n=40, 33, 35, 46, 38) | 1.0 (0.26) | 0.8 (0.16) | 1.0 (0.37) | 1.2 (0.49) | 1.2 (0.32)
  Change from BL to 12 months; (n=37, 29, 30, 41,33) | -0.5 (1.38) | -0.2 (0.42) | 0.1 (0.47) | 0.1 (0.63) | 0.3 (0.33)

18. Secondary Outcome: Mean Change in Baseline Values of Cystatin C at 2 and 12 Months
Description: Cystatin C is a protein encoded by the CST3 gene, which is mainly used as a biomarker of kidney function. If kidney function and glomerular filtration rate decline, the blood levels of cystatin C rise.
Time Frame: Baseline (pretransplant), 2, and 12 months posttransplant
Population: ITT population: all randomized and transplanted participants. n = participants who had both baseline and postbaseline values.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 50 | 48 | 49 | 53 | 50
mg/L
  Baseline (BL); (n=44, 47, 48, 49, 43) | 1.2 (0.64) | 1.2 (0.57) | 1.1 (0.39) | 1.4 (0.73) | 1.2 (0.60)
  2 months; (n=40, 39, 39, 48, 43) | 1.1 (0.26) | 1.1 (0.48) | 1.0 (0.25) | 1.4 (0.52) | 1.5 (0.47)
  Change from BL to 2 months; (n=35, 38, 38, 44,37) | -0.2 (0.62) | -0.1 (0.72) | -0.1 (0.31) | 0.1 (0.77) | 0.3 (0.70)
  12 months; (n=40, 36, 36, 49, 40) | 1.1 (0.36) | 0.9 (0.28) | 1.2 (0.79) | 1.3 (0.53) | 1.3 (0.35)
  Change from BL to 12 months; (n=35, 35, 35,45,34) | -0.2 (0.64) | -0.2 (0.63) | 0.1 (0.86) | -0.1 (0.69) | 0.1 (0.63)

19. Secondary Outcome: Belatacept Pharmacokinetic (PK) Parameter: Maximum Serum Concentration
Description: Maximum Plasma Concentration (Cmax) is the maximum observed serum drug concentration.
Time Frame: Samples were collected at Pre dose on Days 5, 14, 28, 56, 84, 112, 168, 252, 336, 364; after end of infusion on Days 1, 5, 84, 112, 196, 336; and on Days 9, 85, 91, 98, 105.
Population: All randomized participants who received belatacept, and had complete PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 12 | 11 | 11 | 0 | 0
µg/mL | 221.3 (29) | 227.6 (23) | 205.4 (20) |  |

20. Secondary Outcome: Belatacept Pharmacokinetic (PK) Parameter: Time to Achieve the Maximum Plasma Concentration
Description: Maximum Plasma Concentration (Tmax) is the time taken to reach the maximum observed plasma concentration.
Time Frame: as for outcome 19
Population: All randomized participants who received belatacept, and had complete PK profile.
Measure: Median (Full Range); unit: hour
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 12 | 11 | 11 | 0 | 0
hour | 1.00 [0.5 to 1.67] | 1.08 [0.75 to 1.50] | 1.00 [0.83 to 1.17] |  |

21. Secondary Outcome: Belatacept PK Parameter: Area Under the Serum Concentration-time Curve to the End of the Dosing Period (AUCtau)
Description: Area under the plasma concentration-time curve for each dosing interval is determined using the linear trapezoidal rule. The AUC(TAU) of belatacept from the MI regimens and LI regimens were calculated over 2 and 4 weeks respectively.
Time Frame: as for outcome 19
Population: All randomized participants who received belatacept, and had complete PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/mL
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 10 | 5 | 6 | 0 | 0
µg*h/mL | 19865 (21) | 21526 (44) | 19730 (22) |  |

22. Secondary Outcome: Belatacept PK Parameter: Minimum Plasma Concentration
Description: Minimum Plasma Concentration (Cmin) is the minimum observed serum drug concentration.
Time Frame: as for outcome 19
Population: All randomized participants who received belatacept, and had complete PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 13 | 11 | 12 | 0 | 0
µg/mL | 23.63 (30) | 27.20 (37) | 5.91 (50) |  |

23. Secondary Outcome: Belatacept PK Parameter: Terminal Half-life
Description: Terminal Half-life (T 1/2) is the time a drug takes for the concentration levels to fall to 50% of their value.
Time Frame: as for outcome 19
Population: All randomized participants who received belatacept, and had complete PK profile.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 10 | 5 | 7 | 0 | 0
hour | 240.80 (47.82) | 227.74 (56.15) | 207.88 (31.66) |  |

24. Secondary Outcome: Belatacept PK Parameter: Total Body Clearance
Description: Total body clearance is the rate and extent at which the drug is eliminated from the body. The clearance of a drug is used to understand the processes involved in drug elimination, distribution and metabolism. CLT was estimated from AUC (TAU) between Weeks 12 and 16, assuming steady state.
Time Frame: as for outcome 19
Population: All randomized participants who received belatacept, and had complete PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h/kg
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 10 | 5 | 6 | 0 | 0
mL/h/kg | 0.45 (28) | 0.41 (46) | 0.45 (22) |  |

25. Secondary Outcome: Belatacept PK Parameter: Volume of Distribution
Description: Volume of distribution (Vss) is the volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration. . Vss was estimated from AUC (TAU) between Weeks 12 and 16, assuming steady state.
Time Frame: as for outcome 19
Population: All randomized participants who received belatacept, and had complete PK profile.
Measure: Mean (Standard Deviation); unit: L/kg
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 10 | 5 | 6 | 0 | 0
L/kg | 0.09 (0.02) | 0.08 (0.04) | 0.11 (0.03) |  |

26. Secondary Outcome: Belatacept PK Parameter: Amount Excreted in Ascites Fluid Over Days 1 to 14
Description: Amount Excreted in Ascites (Ae,asc) was estimated from the ascites drug concentrations and volumes within a dosing interval.
Time Frame: Days 1 to 14
Population: All randomized participants who received belatacept, and had complete PK profile.
Measure: Mean (Standard Deviation); unit: µg
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 8 | 8 | 12 | 0 | 0
µg | 46654 (59210) | 31425 (40382) | 81451 (95931) |  |

27. Secondary Outcome: Belatacept PK Parameter: Clearance From Ascites Fluid
Description: Clearance from ascites fluid was determined by amount excreted in ascites fluid (Ae, asc)[0-T] / AUC[0-T], where 0-T is the same duration relative to a belatacept infusion.
Time Frame: Days 1 to 14
Population: Serum AUC was not available for the time interval corresponding to ascites fluid collection.
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

28. Secondary Outcome: Belatacept Trough Concentration Before Each Infusion During the LTE
Description: Minimum Plasma Concentration (Cmin) is the minimum observed serum drug concentration.
Time Frame: Samples were collected predose on Days 5, 14, 28, 56, 84, 112, 168, 252, 336, 364; after end of infusion on Days 1, 5, 84, 112, 196, 336; and on Days 9, 85, 91, 98, 105, 532, 728.
Population: All randomized participants who received Belatacept, and had complete PK profile. n= participants with values at all time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 50 | 48 | 49 | 0 | 0
µg/mL
  Day 5: (n=40, 43, 41) | 79.15 (33.32) | 79.40 (33.19) | 70.88 (38.66) |  |
  Day 14: (n=41, 43, 38) | 32.39 (40.85) | 31.16 (39.74) | 29.21 (47.62) |  |
  Day 28: (n=42, 38, 37) | 23.51 (46.71) | 22.23 (47.49) | 21.72 (47.64) |  |
  Day 56: (n=12, 13, 12) | 18.91 (39.74) | 18.84 (36.85) | 6.57 (82.41) |  |
  Day 84: (n=34, 31, 34 ) | 27.11 (38.29) | 27.32 (56.13) | 6.60 (54.25) |  |
  Day 112: (n=29, 26, 29) | 10.12 (63.71) | 9.64 (59.28) | 6.75 (64.11) |  |
  Day 168: (n=30, 29, 29) | 7.30 (58.14) | 8.01 (64.97) | 3.57 (52.56) |  |
  Day 252: (n=28, 28, 27) | 3.65 (67.07) | 3.74 (65.78) | 3.59 (50.93) |  |
  Day 336: (n=26, 23, 21) | 3.22 (70.42) | 3.38 (62.10) | 4.37 (29.72) |  |
  Day 364: (n=28, 28, 22 ) | 2.52 (70.82) | 4.01 (55.68) | 3.62 (48.17) |  |
  Day 532: (n=22, 24, 14) | 2.71 (55.53) | 4.68 (57.61) | 4.91 (34.49) |  |
  Day 728: (n=10, 12, 14) | 4.75 (53.56) | 4.20 (59.28) | 4.22 (46.73) |  |

29. Secondary Outcome: Percentage of Participants (Who Were Hepatitis C Virus [HCV] Positive at Baseline) With HCV Recurrence (Assessed by Central Pathologist) by 12 Months
Description: HCV Recurrence is defined as Histological confirmation on liver biopsy by the Ishak (modified Knodell) system and required both a score >= 5 out of 18 on modified Histological Activity Index grading and a fibrosis Score >= 2 out of 6 on modified staging. All biopsies, including Week 52 biopsies, were considered. Only the first HCV recurrence episode for each participant was counted. For 95% CI within each group, normal approximation was used if N>=5, otherwise exact method was used. For 95% CI of difference, normal approximation was used if N>=5 in both arms, otherwise exact method was used.
Time Frame: 6 and 12 months posttransplant
Population: ITT population, all randomized and transplanted participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Group 1: Basiliximab+Belatacept (MI) + MMF: Basiliximab ; Intravenous (IV), 20 mg, Day 1 and Day 5 Belatacept More Intensive (MI) ; Intravenous (IV), 10 mg/kg on Days 1, 3 and 5, and at Weeks 2, 4, 6, 8, 10, 12, 16, 20, and 24. After 6 months (24 weeks) 5 mg/kg, every 4 weeks, 52 weeks (Short term [ST]), 5 mg/kg, every 4 weeks, 4 years (Long-term extension [LTE]); Mycophenolate Mofetil (MMF), Intravenous (IV)/Capsules, IV/Oral, 1-2g/day, 52 weeks (Short term [ST]), ≤ 1 g/day, 4 years (Long-term extension [LTE])
- Group 2: Belatacept (MI) + MMF: Belatacept More Intensive (MI): IV, 10 mg/kg on Days 1, 3 and 5, and at Weeks 2, 4, 6, 8, 10, 12, 16, 20, and 24. After 6 months (24 weeks) 5 mg/kg, every 4 weeks, 52 weeks (ST), 5 mg/kg, every 4 weeks, 4 years (LTE) + MMF , Intravenous (IV)/Capsules, IV/Oral, 1-2g/day, 52 weeks (ST), ≤ 1 g/day, 4 years (LTE)
- Group 3: Belatacept Less Intensive (LI) + MMF: Drug: Belatacept Less Intensive (LI), IV, 10 mg/kg on Days 1, 3 and 5, and at Weeks 2, 4, 8 and 12. After 3 months (12 weeks) 5 mg/kg, every 4 weeks, 52 weeks (Short term [ST]), 5 mg/kg, every 4 weeks, 4 years (LTE) + MMF, Intravenous (IV)/Capsules, IV/Oral, 1-2g/day, 52 weeks (ST), ≤ 1 g/day, 4 years (LTE)
- Group 4: Tacrolimus + MMF: Tacrolimus, Capsules, Oral, 6-12 ng/mL trough level, twice daily, 52 weeks (Short Term [ST]), in accordance with local practice and the package insert, 4 years (LTE) + MMF, IV/Capsules, IV/Oral, 1-2g/day, 52 weeks (ST), ≤ 1 g/day, 4 years (LTE)
- Group 5: Tacrolimus: Tacrolimus, Capsules, Oral, 6-12 ng/mL trough level, twice daily, 52 weeks (ST), in accordance with local practice and the package insert, 4 years (LTE)
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept Less Intensive (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 23 | 23 | 21 | 25 | 24
percentage of participants
  6 months | 39.1 [19.2 to 59.1] | 21.7 [4.9 to 38.6] | 23.8 [5.6 to 42.0] | 20.0 [4.3 to 35.7] | 33.3 [14.5 to 52.2]
  12 months | 60.9 [40.9 to 80.8] | 30.4 [11.6 to 49.2] | 28.6 [9.2 to 47.9] | 52.0 [32.4 to 71.6] | 37.5 [18.1 to 56.9]
Statistical Analysis 1: Comparison: Group 1: Basiliximab+Belatacept (MI) + MMF vs Group 4: Tacrolimus + MMF; Analysis at Month 6; Test type: Superiority or Other; Mean Difference (Final Values) = 19.1, 95% CI 2-sided [-6.7 to 43.3] — For 95% CI of difference, normal approximation was used if N >= 5 in each treatment arm. Otherwise exact method ignoring stratification was used
Statistical Analysis 2: Comparison: Group 2: Belatacept (MI) + MMF vs Group 4: Tacrolimus + MMF; Analysis at Month 6; Test type: Superiority or Other; Mean Difference (Final Values) = 1.7, 95% CI 2-sided [-21.6 to 25.5] — [estimate comment as in outcome 29, analysis 1]
Statistical Analysis 3: Comparison: Group 3: Belatacept Less Intensive (LI) + MMF vs Group 4: Tacrolimus + MMF; Analysis at Month 6; Test type: Superiority or Other; Mean Difference (Final Values) = 3.8, 95% CI 2-sided [-20.1 to 28.7] — [estimate comment as in outcome 29, analysis 1]
Statistical Analysis 4: Comparison: Group 1: Basiliximab+Belatacept (MI) + MMF vs Group 5: Tacrolimus; Analysis at Month 6; Test type: Superiority or Other; Mean Difference (Final Values) = 5.8, 95% CI 2-sided [-21.2 to 32.1] — [estimate comment as in outcome 29, analysis 1]
Statistical Analysis 5: Comparison: Group 2: Belatacept (MI) + MMF vs Group 5: Tacrolimus; Analysis at Month 6; Test type: Superiority or Other; Mean Difference (Final Values) = -11.6, 95% CI 2-sided [-36.0 to 14.2] — [estimate comment as in outcome 29, analysis 1]
Statistical Analysis 6: Comparison: Group 3: Belatacept Less Intensive (LI) + MMF vs Group 5: Tacrolimus; Analysis at Month 6; Test type: Superiority or Other; Mean Difference (Final Values) = -9.5, 95% CI 2-sided [-34.6 to 17.3] — [estimate comment as in outcome 29, analysis 1]
Statistical Analysis 7: Comparison: Group 1: Basiliximab+Belatacept (MI) + MMF vs Group 4: Tacrolimus + MMF; Analysis at Month 12; Test type: Superiority or Other; Mean Difference (Final Values) = 8.9, 95% CI 2-sided [-18.8 to 35.1] — [estimate comment as in outcome 29, analysis 1]
Statistical Analysis 8: Comparison: Group 2: Belatacept (MI) + MMF vs Group 4: Tacrolimus + MMF; Analysis at Month 12; Test type: Superiority or Other; Mean Difference (Final Values) = -21.6, 95% CI 2-sided [-46.3 to 6.3] — [estimate comment as in outcome 29, analysis 1]
Statistical Analysis 9: Comparison: Group 3: Belatacept Less Intensive (LI) + MMF vs Group 4: Tacrolimus + MMF; Analysis at Month 12; Test type: Superiority or Other; Mean Difference (Final Values) = -23.4, 95% CI 2-sided [-48.2 to 5.2] — [estimate comment as in outcome 29, analysis 1]
Statistical Analysis 10: Comparison: Group 1: Basiliximab+Belatacept (MI) + MMF vs Group 5: Tacrolimus; Analysis at Month 12; Test type: Superiority or Other; Mean Difference (Final Values) = 23.4, 95% CI 2-sided [-5.2 to 48.4] — [estimate comment as in outcome 29, analysis 1]
Statistical Analysis 11: Comparison: Group 2: Belatacept (MI) + MMF vs Group 5: Tacrolimus; Analysis at Month 12; Test type: Superiority or Other; Mean Difference (Final Values) = -7.1, 95% CI 2-sided [-32.9 to 19.8] — [estimate comment as in outcome 29, analysis 1]
Statistical Analysis 12: Comparison: Group 3: Belatacept Less Intensive (LI) + MMF vs Group 5: Tacrolimus; Analysis at Month 12; Test type: Superiority or Other; Mean Difference (Final Values) = -8.9, 95% CI 2-sided [-34.8 to 18.7] — [estimate comment as in outcome 29, analysis 1]

30. Secondary Outcome: Percentage of Participants (Who Were Hepatitis C Virus [HCV] Positive at Baseline) With HCV Recurrence (Assessed by Central Pathologist) During the LTE
Description: as for outcome 29
Time Frame: 12 months posttransplant, end of study (database lock, 20-June-2011)
Population: ITT-LTE population, all randomized and transplanted participants who entered long-term extension.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept Less Intensive (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 12 | 12 | 9 | 17 | 11
percentage of participants
  At 12 months | 50.0 [21.7 to 78.3] | 41.7 [13.8 to 69.6] | 0 [NA to NA] — Not applicable as no subjects had HCV recurrence | 58.8 [35.4 to 82.2] | 72.7 [46.4 to 99.0]
  At end of study | 66.7 [40.0 to 93.3] | 50.0 [21.7 to 78.3] | 22.2 [2.8 to 60.0] | 64.7 [42.0 to 87.4] | 72.7 [46.4 to 99.0]
Statistical Analysis 1: Comparison: Group 1: Basiliximab+Belatacept (MI) + MMF vs Group 4: Tacrolimus + MMF; Analysis at Month 12; Test type: Superiority or Other; Mean Difference (Final Values) = -8.8, 95% CI 2-sided [-42.4 to 26.3] — For 95% CI of difference, normal approximation was used if N >= 5 in each treatment arm. Otherwise exact method was used
Statistical Analysis 2: Comparison: Group 2: Belatacept (MI) + MMF vs Group 4: Tacrolimus + MMF; Analysis at Month 12; Test type: Superiority or Other; Mean Difference (Final Values) = -17.2, 95% CI 2-sided [-49.2 to 19.0] — [estimate comment as in outcome 30, analysis 1]
Statistical Analysis 3: Comparison: Group 3: Belatacept Less Intensive (LI) + MMF vs Group 4: Tacrolimus + MMF; Analysis at Month 12; Test type: Superiority or Other; Mean Difference (Final Values) = -58.8, 95% CI 2-sided [-81.6 to -19.8] — [estimate comment as in outcome 30, analysis 1]
Statistical Analysis 4: Comparison: Group 1: Basiliximab+Belatacept (MI) + MMF vs Group 5: Tacrolimus; Analysis at Month 12; Test type: Superiority or Other; Mean Difference (Final Values) = -22.7, 95% CI 2-sided [-55.9 to 16.9] — [estimate comment as in outcome 30, analysis 1]
Statistical Analysis 5: Comparison: Group 2: Belatacept (MI) + MMF vs Group 5: Tacrolimus; Analysis at Month 12; Test type: Superiority or Other; Mean Difference (Final Values) = -31.1, 95% CI 2-sided [-62.6 to 9.4] — [estimate comment as in outcome 30, analysis 1]
Statistical Analysis 6: Comparison: Group 3: Belatacept Less Intensive (LI) + MMF vs Group 5: Tacrolimus; Analysis at Month 12; Test type: Superiority or Other; Mean Difference (Final Values) = -72.7, 95% CI 2-sided [-94.0 to -33.1] — [estimate comment as in outcome 30, analysis 1]
Statistical Analysis 7: Comparison: Group 1: Basiliximab+Belatacept (MI) + MMF vs Group 4: Tacrolimus + MMF; Analysis at database lock; Test type: Superiority or Other; Mean Difference (Final Values) = 2.0, 95% CI 2-sided [-32.6 to 34.3] — [estimate comment as in outcome 30, analysis 1]
Statistical Analysis 8: Comparison: Group 2: Belatacept (MI) + MMF vs Group 4: Tacrolimus + MMF; Analysis at database lock; Test type: Superiority or Other; Mean Difference (Final Values) = -14.7, 95% CI 2-sided [-47.4 to 20.6] — [estimate comment as in outcome 30, analysis 1]
Statistical Analysis 9: Comparison: Group 3: Belatacept Less Intensive (LI) + MMF vs Group 4: Tacrolimus + MMF; Analysis at database lock; Test type: Superiority or Other; Mean Difference (Final Values) = -42.5, 95% CI 2-sided [-72.6 to 0.5] — [estimate comment as in outcome 30, analysis 1]
Statistical Analysis 10: Comparison: Group 1: Basiliximab+Belatacept (MI) + MMF vs Group 5: Tacrolimus; Analysis at database lock; Test type: Superiority or Other; Mean Difference (Final Values) = -6.1, 95% CI 2-sided [-41.1 to 31.1] — [estimate comment as in outcome 30, analysis 1]
Statistical Analysis 11: Comparison: Group 2: Belatacept (MI) + MMF vs Group 5: Tacrolimus; Analysis at database lock; Test type: Superiority or Other; Mean Difference (Final Values) = -22.7, 95% CI 2-sided [-55.9 to 16.9] — [estimate comment as in outcome 30, analysis 1]
Statistical Analysis 12: Comparison: Group 3: Belatacept Less Intensive (LI) + MMF vs Group 5: Tacrolimus; Analysis at database lock; Test type: Superiority or Other; Mean Difference (Final Values) = -50.5, 95% CI 2-sided [-81.9 to -3.5] — [estimate comment as in outcome 30, analysis 1]

31. Secondary Outcome: Number of Participants (Who Were HCV Positive at Baseline) With HCV Ribonucleic Acid (RNA) Levels >2.4*10^6 U/mL and >4.7*10^6 U/mL: 12-month Treatment Phase
Description: Recurrent hepatitis C infection of the allograft following liver transplantation can be detected by monitoring HCV RNA levels. In HCV positive participants, quantitative HCV RNA levels > 2.4 * 10^6 U/mL and > 4.7 * 10^6 U/mL were descriptively summarized by treatment group. BL=baseline
Time Frame: Baseline (pretransplant), 6 and 12 months (mo) posttransplant
Population: ITT population, all randomized and transplanted participants. n= participants who were HCV positive at baseline.
Measure: Number; unit: participants
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept Less Intensive (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 23 | 23 | 21 | 25 | 24
participants
  BL; HCV RNA > 2.4*10^6 U/mL (n=21,22,19,22,23) | 2 | 4 | 2 | 3 | 1
  BL; HCV RNA > 4.7 *10^6 U/mL (n=21,22,19,22,23) | 0 | 1 | 1 | 0 | 0
  6 mo; HCV RNA > 2.4*10^6 U/mL (n=16,15,15,21,14) | 9 | 7 | 8 | 14 | 11
  6 mo; HCV RNA > 4.7*10^6 U/mL (n=16,15,15,21,14) | 7 | 7 | 7 | 11 | 10
  12 mo; HCV RNA > 2.4*10^6 U/mL (n=15,13,14,20,13) | 7 | 7 | 7 | 13 | 7
  12 mo; HCV RNA > 4.7*10^6 U/mL (n=15,13,14,20,13) | 6 | 6 | 5 | 11 | 7

32. Secondary Outcome: Number of Participants (Who Were HCV Positive at Baseline) With HCV RNA Levels >2.4 * 10^6 U/mL and >4.7 * 10^6 U/mL During the LTE
Description: Recurrent hepatitis C infection of the allograft following liver transplantation can be detected by monitoring HCV RNA levels. In HCV positive participants, quantitative HCV RNA levels > 2.4 x 10^6 U/mL and > 4.7 x 10^6 U/mL were descriptively summarized by treatment group. BL = baseline
Time Frame: BL (pretransplant), 12, 18, 24, 30 months (mo) posttransplant
Population: ITT-LTE population, all randomized and transplanted participants. n= participants with HCV RNA values.
Measure: Number; unit: participants
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept Less Intensive (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 12 | 12 | 9 | 17 | 11
participants
  BL; HCV RNA > 2.4*10^6 U/mL (n=10,11,6,15,10) | 0 | 1 | 0 | 2 | 1
  12 mo; HCV RNA > 2.4*10^6 U/mL (n=11,10,8,16,10) | 6 | 5 | 4 | 10 | 4
  12 mo; HCV RNA > 4.7*10^6 U/mL (n=11,10,8,16,10) | 6 | 4 | 3 | 8 | 4
  18 mo; HCV RNA > 2.4*10^6 U/mL (n=7,10,3,12,9) | 3 | 2 | 2 | 7 | 3
  18 mo; HCV RNA > 4.7*10^6 U/mL (n=7,10,3,12,9) | 2 | 2 | 2 | 6 | 2
  24 mo; HCV RNA > 2.4*10^6 U/mL (n=4,3,4,8,4) | 2 | 1 | 1 | 6 | 1
  24 mo; HCV RNA > 4.7*10^6 U/mL (n=4,3,4,8,4) | 2 | 0 | 0 | 5 | 1
  30 mo; HCV RNA > 2.4*10^6 U/mL (n=1,1,1,2,2) | 1 | 0 | 0 | 1 | 1
  30 mo; HCV RNA > 4.7*10^6 U/mL (n=1,1,1,2,2) | 1 | 0 | 0 | 1 | 1

33. Secondary Outcome: Percentage of Participants Who Develop Dyslipidemia, Hypertriglyceridemia and Hypercholesterolemia After Randomization and Transplantation: 12-month Treatment Phase
Description: Percentage of participants who develop dyslipidemia, defined as hypertriglyceridemia (triglycerides [TGs] ≥ 500 mg/dL [5.65 mmol/L]), hypercholesterolemia (Low density lipoprotein [LDL] ≥ 100 mg/dL [2.59 mmol/L]), or elevated non-high density lipoprotein (non- high density lipoprotein [HDL] ≥ 130 mg/dL [3.36 mmol/L]) in the presence of high TGs (TGs ≥ 200 mg/dL [2.26 mmol/L]).
Time Frame: 6 and 12 months posttransplant
Population: ITT population, all randomized and transplanted participants who did not have dyslipidemia at baseline
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept Less Intensive (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 42 | 35 | 46 | 42 | 37
percentage of participants
  By 6 month: Dyslipidemia | 50.0 [34.9 to 65.1] | 54.3 [37.8 to 70.8] | 45.7 [31.3 to 60.0] | 33.3 [19.1 to 47.6] | 59.5 [43.6 to 75.3]
  By 6 month: Hypertriglyceridemia | 2.4 [0.1 to 12.6] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  By 6 month: Hypercholesterolemia | 42.9 [27.9 to 57.8] | 48.6 [32.0 to 65.1] | 39.1 [25.0 to 53.2] | 28.6 [14.9 to 42.2] | 51.4 [35.2 to 67.5]
  By 12 month: Dyslipidemia | 59.5 [44.7 to 74.4] | 57.1 [40.7 to 73.5] | 58.7 [44.5 to 72.9] | 50.0 [34.9 to 65.1] | 70.3 [55.5 to 85.0]
  By 12 month: Hypertriglyceridemia | 4.8 [0.6 to 16.2] | 0 [0 to 0] | 2.2 [0.1 to 11.5] | 2.4 [0.1 to 12.6] | 0 [0 to 0]
  By 12 month: Hypercholesterolemia | 54.8 [39.7 to 69.8] | 54.3 [37.8 to 70.8] | 52.2 [37.7 to 66.6] | 42.9 [27.9 to 57.8] | 62.2 [46.5 to 77.8]

34. Secondary Outcome: Percentage of Participants Meeting the Definition of Dyslipidemia, Hypertriglyceridemia or Hypercholesterolemia at Any Given Time: 12-month Treatment Phase
Description: Percentage of participants at any given time (at Month 6 and Month 12) who met the definition of dyslipidemia.Dyslipidemia is defined as hypertriglyceridemia (TGs ≥ 500 mg/dL [5.65 mmol/L]), hypercholesterolemia (LDL ≥ 100 mg/dL [2.59 mmol/L]), or elevated non-HDL (non-HDL ≥ 130 mg/dL [3.36 mmol/L]) in the presence of high TGs (TGs ≥ 200 mg/dL [2.26 mmol/L]).
Time Frame: 6 and 12 months posttransplant
Population: ITT population, all randomized and transplanted participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept Less Intensive (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 50 | 48 | 49 | 53 | 50
percentage of participants
  6 months: Dyslipidemia | 36.0 [22.7 to 49.3] | 31.3 [18.1 to 44.4] | 30.6 [17.7 to 43.5] | 32.1 [19.5 to 44.6] | 26.0 [13.8 to 38.2]
  6 months: Hypertriglyceridemia | 6.0 [1.3 to 16.5] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  6 months: Hypercholesterolemia | 30.0 [17.3 to 42.7] | 29.2 [16.3 to 42.0] | 24.5 [12.4 to 36.5] | 30.2 [17.8 to 42.5] | 22.0 [10.5 to 33.5]
  12 months: Dyslipidemia | 40.0 [26.4 to 53.6] | 33.3 [20.0 to 46.7] | 44.9 [31.0 to 58.8] | 34.0 [21.2 to 46.7] | 42.0 [28.3 to 55.7]
  12 months: Hypertriglyceridemia | 4.0 [0.5 to 13.7] | 0 [0 to 0] | 2.0 [0.1 to 10.9] | 1.9 [0.0 to 10.1] | 2.0 [0.1 to 10.6]
  12 months: Hypercholesterolemia | 30.0 [17.3 to 42.7] | 29.2 [16.3 to 42.0] | 40.8 [27.1 to 54.6] | 30.2 [17.8 to 42.5] | 36.0 [22.7 to 49.3]

35. Secondary Outcome: Summary Statistics for Lipid Parameters-Serum Total Non-High Density Lipoprotein (Non-HDL) Cholesterol: 12-month Treatment Phase
Time Frame: Baseline (pretransplant), 1, 6, 12 months posttransplant
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept Less Intensive (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 50 | 48 | 49 | 53 | 50
mg/dL
  BL (n=45, 42, 44, 49, 46) | 80.4 (37.1) | 83.5 (44.2) | 84.8 (60.76) | 77.7 (44.30) | 76.8 (46.85)
  1 months (n=46, 47, 42, 49, 49) | 125.1 (42.91) | 147.9 (82.96) | 148.0 (71.11) | 121.7 (40.25) | 130.0 (50.75)
  Change from BL to 1 months (n=42, 41, 39, 45, 45) | 47.2 (50.14) | 66.0 (102.0) | 54.1 (86.63) | 47.0 (61.36) | 47.5 (50.32)
  6 months (n=39, 34, 38, 48, 36) | 139.3 (48.93) | 134.4 (45.16) | 138.9 (43.39) | 125.1 (44.02) | 135.4 (58.49)
  Change from BL to 6 months (n=35, 30, 35, 44, 32) | 59.5 (48.06) | 44.0 (54.37) | 48.2 (75.74) | 48.1 (51.09) | 48.6 (76.78)
  12 months (n=40, 33, 35, 45, 37) | 143.2 (84.77) | 137.4 (38.49) | 142.2 (62.41) | 118.2 (43.00) | 131.9 (39.71)
  Change from BL to 12 months (n=35, 29, 32, 42, 33) | 66.7 (80.64) | 49.2 (63.87) | 53.4 (97.28) | 47.4 (54.80) | 44.1 (72.35)

36. Secondary Outcome: Summary Statistics for Lipid Parameters; Serum HDL Cholesterol: 12-month Treatment Phase
Time Frame: Baseline (pretransplant), 1, 6, 12 months posttransplant
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept Less Intensive (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 50 | 48 | 49 | 53 | 50
mg/dL
  BL (n=46, 42, 44, 49, 46) | 32.1 (17.38) | 36.2 (17.49) | 36.5 (19.66) | 33.3 (21.97) | 31.1 (15.50)
  1 month (n=46, 47, 42, 49, 49) | 41.3 (15.37) | 36.9 (17.80) | 42.5 (19.60) | 41.2 (11.32) | 34.1 (14.11)
  Change from BL to 1month (n=43, 41, 39, 45, 45) | 9.9 (26.83) | 1.7 (26.15) | 7.2 (27.72) | 7.1 (22.65) | 3.4 (21.37)
  6 months (n=39, 34, 38, 48, 36) | 41.5 (14.29) | 42.8 (14.17) | 44.2 (14.56) | 45.5 (15.80) | 42.6 (17.92)
  Change from BL to 6 months (n=36, 30, 35, 44, 32) | 9.2 (21.56) | 7.3 (20.40) | 9.4 (22.06) | 10.8 (28.26) | 9.5 (24.32)
  12 months (n=40, 33, 35, 45, 37) | 43.6 (14.40) | 41.5 (15.19) | 44.2 (14.37) | 45.6 (15.35) | 43.3 (15.58)
  Change from BL to12 months (n=36, 29, 32, 42, 33) | 12.7 (23.25) | 8.3 (22.75) | 7.3 (24.71) | 10.9 (24.13) | 10.0 (21.01)

37. Secondary Outcome: Summary Statistics for Lipid Parameters- Serum Low Density Lipoprotein Cholesterol (LDL): 12-month Treatment Phase
Time Frame: Baseline (pretransplant), 1, 6, 12 months posttransplant
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept Less Intensive (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 50 | 48 | 49 | 53 | 50
mg/dL
  BL (n=29, 30, 25, 34, 32) | 52.3 (25.26) | 58.6 (34.97) | 58.9 (34.08) | 63.6 (45.02) | 59.9 (42.60)
  1 month (n=30, 34, 29, 41, 42) | 95.2 (33.82) | 93.2 (33.73) | 115.7 (58.88) | 89.8 (37.31) | 98.4 (47.68)
  Change from BL to 1 month (n=17, 21, 17, 27, 30) | 42.7 (47.94) | 34.3 (48.98) | 57.1 (30.19) | 26.1 (48.40) | 41.5 (43.68)
  6 months (n=27, 29, 27, 41, 30) | 99.2 (36.93) | 107.5 (36.93) | 98.2 (42.85) | 96.7 (42.22) | 92.8 (29.03)
  Change from BL to 6 months (n=16, 19, 18, 28, 22) | 41.2 (33.82) | 45.9 (42.13) | 48.7 (41.66) | 28.9 (49.29) | 26.1 (54.04)
  12 months (n=38, 29, 32, 42, 35) | 93.0 (30.72) | 107.2 (32.75) | 103.2 (36.41) | 89.0 (37.15) | 93.8 (27.45)
  Change from BL to 12 months (n=22, 19, 20, 25, 22) | 37.8 (33.09) | 45.4 (51.75) | 37.2 (47.81) | 23.7 (46.80) | 13.7 (50.98)

38. Secondary Outcome: Summary Statistics for Lipid Parameters- Serum Cholesterol: 12-month Treatment Phase
Time Frame: Baseline (pretransplant), 1, 6, 12 months posttransplant
Population: ITT population, all randomized and transplanted participants.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept Less Intensive (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 50 | 48 | 49 | 53 | 50
mg/dL
  BL (n=45, 42, 44, 49, 47) | 112.9 (49.76) | 119.7 (51.81) | 121.3 (63.05) | 111.0 (54.91) | 106.4 (51.82)
  1 month (n=46, 47, 42, 49, 49) | 166.3 (45.92) | 184.9 (77.16) | 190.6 (69.54) | 162.9 (43.72) | 164.1 (52.95)
  Change from BL to 1 month (n=42, 41, 39, 45, 46) | 57.0 (63.06) | 67.7 (102.3) | 61.3 (84.20) | 54.0 (70.01) | 53.4 (57.19)
  6 months (n=39, 34, 38, 48, 36) | 180.8 (52.76) | 177.3 (49.56) | 182.2 (45.58) | 170.6 (49.30) | 177.9 (57.92)
  Change from BL to 6 months (n=35, 30, 35, 44, 33) | 68.6 (60.07) | 51.3 (63.22) | 56.6 (72.89) | 58.9 (66.3) | 60.8 (71.33)
  12 months (n=40, 33, 35, 45, 37) | 186.8 (87.16) | 178.9 (42.13) | 186.4 (59.11) | 163.8 (46.41) | 175.2 (38.37)
  Change from BL to 12 months (n=35, 29,32, 42, 34) | 79.4 (86.88) | 57.5 (73.67) | 60.7 (92.87) | 58.2 (64.05) | 57.3 (72.22)

39. Secondary Outcome: Summary Statistics for Lipid Parameters - Serum Triglyceride: 12-month Treatment Phase
Time Frame: Baseline (pretransplant), 1, 6, 12 months posttransplant
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept Less Intensive (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 50 | 48 | 49 | 53 | 50
mg/dL
  BL (n=29, 30, 25, 34, 32) | 94.4 (60.42) | 110.1 (135.1) | 80.2 (46.29) | 84.4 (34.22) | 89.2 (73.45)
  1 month (n=29, 33, 29, 41, 43) | 153.9 (65.83) | 162.9 (108.1) | 149.0 (72.84) | 149.1 (61.27) | 163.5 (73.80)
  Change from BL to 1 month (n=16, 20, 17, 27, 30) | 71.2 (84.87) | 45.7 (223.0) | 85.8 (93.63) | 68.2 (75.45) | 71.8 (58.66)
  6 months (n=26, 29, 25, 41, 30) | 234.3 (316.6) | 157.1 (82.23) | 162.7 (109.2) | 148.1 (67.50) | 167.2 (100.8)
  Change from BL to 6 months (n=15, 19, 18, 28, 22) | 199.9 (329.1) | 18.3 (140.8) | 88.7 (113.1) | 60.8 (63.06) | 84.3 (105.2)
  12 months (n=38, 29, 32, 42, 34) | 255.1 (582.7) | 159.0 (70.77) | 158.2 (99.93) | 156.4 (105.7) | 190.5 (125.7)
  Change from BL to 12 months (n=22, 19, 20, 25, 21) | 237.2 (703.9) | 20.3 (180.9) | 91.6 (118.0) | 72.3 (60.61) | 92.6 (116.4)

40. Secondary Outcome: Summary Statistics for Systolic Blood Pressure: 12-month Treatment Phase
Time Frame: Baseline (pretransplant), 1, 3, 6, 9, 12 months posttransplant
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept Less Intensive (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 50 | 48 | 49 | 53 | 50
mm Hg
  BL (n=50, 48, 49, 53, 49) | 115.3 (18.41) | 115.4 (22.35) | 111.4 (15.80) | 121.2 (17.31) | 125.3 (21.87)
  1 month (n=50, 48, 49, 52, 48) | 123.3 (16.87) | 126.3 (15.44) | 120.9 (16.96) | 129.2 (13.79) | 124.6 (16.41)
  Change from BL to 1 month (n=50, 48, 49, 52, 47) | 8.0 (19.95) | 10.9 (27.03) | 9.4 (21.65) | 8.5 (18.43) | 0.6 (24.26)
  3 months (n=44, 46, 41, 48, 42) | 127.0 (15.04) | 126.9 (15.03) | 124.4 (17.65) | 136.9 (18.61) | 133.0 (16.18)
  Change from BL to 3 months (n=44, 46, 41, 48, 41) | 10.9 (23.10) | 11.7 (23.85) | 12.7 (21.30) | 16.3 (24.64) | 9.1 (24.99)
  6 months (n=43, 40, 36, 47, 37) | 124.0 (16.09) | 126.5 (15.87) | 124.6 (14.75) | 130.6 (23.29) | 132.0 (22.11)
  Change from BL to 6 months (n=43, 40, 36, 47, 36) | 8.4 (23.18) | 9.3 (24.44) | 12.8 (19.77) | 10.0 (26.62) | 8.3 (27.45)
  9 months (n=34, 30, 29, 41, 31) | 125.5 (16.24) | 125.8 (13.16) | 123.9 (12.22) | 135.6 (20.81) | 133.9 (15.58)
  Change from BL to 9 months (n=34, 30, 29, 41, 31) | 10.4 (21.36) | 8.8 (29.71) | 13.3 (21.94) | 14.4 (26.73) | 11.6 (20.39)
  12 months (n=42, 37, 36, 46, 38) | 125.8 (12.79) | 127.0 (17.02) | 121.2 (13.06) | 137.0 (18.09) | 138.0 (18.67)
  Change from BL to 12 months (n=42, 37, 36, 46, 37) | 9.2 (22.96) | 10.2 (27.33) | 10.6 (17.46) | 15.9 (25.60) | 14.6 (25.88)

41. Secondary Outcome: Summary Statistics for Diastolic Blood Pressure: 12-month Treatment Phase
Description: Participants were considered to have hypertension if they had Diastolic Blood Pressure (SBP) ≥ 80 mmHg.
Time Frame: BL (pretransplant), 1, 3, 6, 9, 12 months posttransplant
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept Less Intensive (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 50 | 48 | 49 | 53 | 50
mm Hg
  BL (n=50, 48, 49, 53, 49) | 64.5 (12.86) | 63.1 (11.50) | 62.9 (10.54) | 67.5 (12.55) | 68.6 (12.07)
  1 month (n=50, 48, 49, 52, 48) | 74.4 (10.34) | 74.7 (9.51) | 72.6 (13.84) | 77.8 (10.26) | 74.6 (10.76)
  Change from BL to 1 month (n=50, 48, 49, 52, 47) | 10.0 (14.53) | 11.7 (12.48) | 9.7 (16.27) | 10.7 (13.80) | 5.8 (14.05)
  3 months (n=44, 46, 41, 48, 42) | 77.4 (9.57) | 78.3 (10.85) | 76.1 (10.81) | 81.7 (10.94) | 78.2 (9.86)
  Change from BL to 3 months (n=44, 46, 41, 48, 41) | 11.5 (14.32) | 15.2 (11.90) | 12.0 (15.70) | 14.4 (15.27) | 9.9 (15.35)
  6 months (n=43, 40, 36, 47, 37) | 74.4 (10.63) | 79.4 (10.17) | 76.3 (9.69) | 77.8 (12.68) | 76.6 (9.11)
  Change from BL to 6 months (n=43, 40, 36, 47, 36) | 8.8 (15.49) | 17.0 (12.86) | 12.5 (14.93) | 10.7 (14.44) | 8.6 (14.58)
  9 months (n=34, 30, 29, 41, 31) | 75.4 (9.96) | 78.5 (11.45) | 77.6 (9.10) | 79.5 (10.74) | 79.5 (10.15)
  Change from BL to 9 months (n=34, 30, 29, 41, 31) | 10.0 (14.41) | 15.2 (16.91) | 13.2 (14.54) | 11.2 (15.37) | 11.2 (13.25)
  12 months (n=42, 37, 36, 46, 38) | 76.5 (9.38) | 78.5 (11.43) | 74.5 (8.54) | 80.3 (10.21) | 79.5 (11.24)
  Change from BL to 12 months (n=42, 37, 36, 46, 37) | 10.26 (15.71) | 16.3 (15.28) | 10.6 (14.35) | 10.21 (13.6) | 10.8 (13.20)

42. Secondary Outcome: Summary Statistics for Mean Arterial Pressure: 12-month Treatment Phase
Time Frame: BL (pretransplant), 1, 3, 6, 9, 12 months posttransplant
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept Less Intensive (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 50 | 48 | 49 | 53 | 50
mm Hg
  BL (n=50, 48, 49, 53, 49) | 81.4 (12.98) | 80.5 (13.58) | 79.1 (10.32) | 85.4 (12.97) | 87.5 (13.42)
  1 month (n=50, 48, 49, 52, 48) | 90.7 (10.97) | 91.9 (10.44) | 88.7 (14.09) | 95.0 (9.89) | 91.3 (11.61)
  Change from BL to 1 month (n=50, 48, 49, 52, 47) | 9.3 (14.58) | 11.4 (14.96) | 9.6 (16.75) | 10.0 (13.86) | 4.1 (15.76)
  3 months (n=44, 46, 41, 48, 41) | 93.9 (9.78) | 94.5 (11.14) | 92.2 (12.18) | 100.1 (12.29) | 96.5 (9.01)
  Change from BL to 3 months (n=44, 46, 41, 48, 41) | 11.3 (15.40) | 14.0 (14.21) | 12.2 (15.95) | 15.1 (17.11) | 9.6 (15.59)
  6 months (n=43, 40, 36, 47, 37) | 91.0 (10.70) | 95.1 (10.92) | 92.4 (9.94) | 95.4 (15.04) | 95.0 (11.70)
  Change from BL to 6 months (n=43, 40, 36, 47, 36) | 8.7 (15.71) | 14.4 (15.63) | 12.6 (14.35) | 10.5 (17.18) | 8.5 (16.74)
  9 months (n=34, 30, 29, 41, 31) | 92.1 (10.41) | 94.3 (10.22) | 93.0 (8.68) | 98.2 (12.46) | 97.7 (10.34)
  Change from BL to 9 months (n=34, 30, 29, 41, 31) | 10.1 (15.06) | 13.1 (19.90) | 13.2 (13.82) | 12.3 (17.71) | 11.3 (13.25)
  12 months (n=42, 37, 36, 46, 38) | 93.0 (8.61) | 94.6 (11.90) | 90.1 (8.89) | 99.2 (11.56) | 99.0 (12.13)
  Change from BL to 12 months (n=42, 37, 36, 46, 37) | 10.1 (15.41) | 14.3 (18.11) | 10.6 (13.06) | 14.3 (17.12) | 12.1 (15.76)

43. Secondary Outcome: Percentage of Participants Who Developed Hypertension in 12-month Treatment Phase
Description: Percentage of participants who develop hypertension after randomization and transplantation. Transient post-operative increases in BP were not to be counted as new onset hypertension. Hypertension was to be assessed only at or after the Week 4 visit. Participants were considered to have hypertension when either of the following criteria were met: (1) SBP ≥ 130 mm Hg or DBP ≥ 80 mm Hg or (2) participant received an antihypertensive medication(s) for the indication of hypertension or due to medical history of hypertension.
Time Frame: 6 and 12 months posttransplant
Population: ITT population, all randomized and transplanted participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept Less Intensive (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 17 | 15 | 16 | 16 | 12
percentage of participants
  By 6 months | 94.1 [82.9 to 100.0] | 93.3 [80.7 to 100.0] | 93.8 [81.9 to 100] | 100.0 [NA to NA] — All the respondents had hypertension, hence CI was not evaluable. | 100 [NA to NA] — All the respondents had hypertension, hence CI was not evaluable.
  By 12 months | 100 [NA to NA] — All the respondents had hypertension, hence confidence interval (CI) not available. | 93.3 [80.7 to 100] | 93.8 [81.9 to 100.0] | 100.0 [NA to NA] — All the respondents had hypertension, hence CI not evaluable. | 100.0 [NA to NA] — All the respondents had hypertension, hence CI not evaluable.
Statistical Analysis 1: Comparison: Group 1: Basiliximab+Belatacept (MI) + MMF vs Group 4: Tacrolimus + MMF; Analysis at Month 6; Test type: Superiority or Other; Mean Difference (Final Values) = -5.9, 95% CI 2-sided [-21.2 to 6.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Group 2: Belatacept (MI) + MMF vs Group 4: Tacrolimus + MMF; Analysis at Month 6; Test type: Superiority or Other; Mean Difference (Final Values) = -6.7, 95% CI 2-sided [-18.2 to 5.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Group 3: Belatacept Less Intensive (LI) + MMF vs Group 4: Tacrolimus + MMF; Analysis at Month 6; Test type: Superiority or Other; Mean Difference (Final Values) = -6.3, 95% CI 2-sided [-14.9 to 4.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Group 1: Basiliximab+Belatacept (MI) + MMF vs Group 5: Tacrolimus; Analysis at Month 6; Test type: Superiority or Other; Mean Difference (Final Values) = -5.9, 95% CI 2-sided [-25.1 to 7.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Group 2: Belatacept (MI) + MMF vs Group 5: Tacrolimus; Analysis at Month 6; Test type: Superiority or Other; Mean Difference (Final Values) = -6.7, 95% CI 2-sided [-15.6 to 4.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Group 3: Belatacept Less Intensive (LI) + MMF vs Group 5: Tacrolimus; Analysis at Month 6; Test type: Superiority or Other; Mean Difference (Final Values) = -6.3, 95% CI 2-sided [-12.7 to 3.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Group 1: Basiliximab+Belatacept (MI) + MMF vs Group 4: Tacrolimus + MMF; Analysis at Month 12; Test type: Superiority or Other; Mean Difference (Final Values) = 0 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Group 2: Belatacept (MI) + MMF vs Group 4: Tacrolimus + MMF; Analysis at Month 12; Test type: Superiority or Other; Mean Difference (Final Values) = -6.7, 95% CI 2-sided [-18.2 to 5.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Group 3: Belatacept Less Intensive (LI) + MMF vs Group 4: Tacrolimus + MMF; Analysis at Month 12; Test type: Superiority or Other; Mean Difference (Final Values) = -6.3, 95% CI 2-sided [-14.9 to 4.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Group 1: Basiliximab+Belatacept (MI) + MMF vs Group 5: Tacrolimus; Analysis at Month 12; Test type: Superiority or Other; Mean Difference (Final Values) = 0 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Group 2: Belatacept (MI) + MMF vs Group 5: Tacrolimus; Analysis at Month 12; Test type: Superiority or Other; Mean Difference (Final Values) = -6.7, 95% CI 2-sided [-15.6 to 4.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Group 3: Belatacept Less Intensive (LI) + MMF vs Group 5: Tacrolimus; Analysis at Month 12; Test type: Superiority or Other; Mean Difference (Final Values) = -6.3, 95% CI 2-sided [-12.7 to 3.9] — [estimate comment as in outcome 1, analysis 1]

44. Secondary Outcome: Percentage of Participants Who Have Hypertension at Any Given Time During the 12-month Treatment Phase
Description: Percentage of participants at any given time who meet the definition of hypertension. Participants were considered to have hypertension when either of the following criteria were met: (1) SBP ≥ 130 mm Hg or DBP ≥ 80 mm Hg or (2) participant received an antihypertensive medication(s) for the indication of hypertension or due to medical history of hypertension.
Time Frame: 6 and 12 months posttransplant
Population: ITT population, all randomized and transplanted participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept Less Intensive (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 50 | 48 | 49 | 53 | 50
percentage of participants
  By 6 months | 64.0 [50.7 to 77.3] | 77.1 [65.2 to 89.0] | 69.4 [56.5 to 82.3] | 71.7 [59.6 to 83.8] | 70.0 [57.3 to 82.7]
  By 12 months | 72.0 [59.6 to 84.4] | 68.8 [55.6 to 81.9] | 59.2 [45.4 to 72.9] | 79.2 [68.3 to 90.2] | 70.0 [57.3 to 82.7]
Statistical Analysis 1: Comparison: Group 1: Basiliximab+Belatacept (MI) + MMF vs Group 4: Tacrolimus + MMF; Analysis at Month 6; Test type: Superiority or Other; Mean Difference (Final Values) = -7.7, 95% CI 2-sided [-25.6 to 10.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Group 2: Belatacept (MI) + MMF vs Group 4: Tacrolimus + MMF; Analysis at Month 6; Test type: Superiority or Other; Mean Difference (Final Values) = 5.4, 95% CI 2-sided [-11.7 to 22.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Group 3: Belatacept Less Intensive (LI) + MMF vs Group 4: Tacrolimus + MMF; Analysis at Month 6; Test type: Superiority or Other; Mean Difference (Final Values) = -2.3, 95% CI 2-sided [-20.1 to 15.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Group 1: Basiliximab+Belatacept (MI) + MMF vs Group 5: Tacrolimus; Analysis at Month 12; Test type: Superiority or Other; Mean Difference (Final Values) = -6.0, 95% CI 2-sided [-24.0 to 12.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Group 2: Belatacept (MI) + MMF vs Group 5: Tacrolimus; Analysis at Month 6; Test type: Superiority or Other; Mean Difference (Final Values) = 7.1, 95% CI 2-sided [-10.5 to 24.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Group 3: Belatacept Less Intensive (LI) + MMF vs Group 5: Tacrolimus; Analysis at Month 6; Test type: Superiority or Other; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-18.5 to 17.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Group 1: Basiliximab+Belatacept (MI) + MMF vs Group 4: Tacrolimus + MMF; Analysis at Month 12; Test type: Superiority or Other; Mean Difference (Final Values) = -7.2, 95% CI 2-sided [-23.3 to 9.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Group 2: Belatacept (MI) + MMF vs Group 4: Tacrolimus + MMF; Analysis at Month 12; Test type: Superiority or Other; Mean Difference (Final Values) = -10.5, 95% CI 2-sided [-27.4 to 6.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Group 3: Belatacept Less Intensive (LI) + MMF vs Group 4: Tacrolimus + MMF; Analysis at Month 12; Test type: Superiority or Other; Mean Difference (Final Values) = -20.1, 95% CI 2-sided [-37.5 to -2.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Group 1: Basiliximab+Belatacept (MI) + MMF vs Group 5: Tacrolimus; Analysis at Month 12; Test type: Superiority or Other; Mean Difference (Final Values) = 2.0, 95% CI 2-sided [-15.5 to 19.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Group 2: Belatacept (MI) + MMF vs Group 5: Tacrolimus; Analysis at Month 12; Test type: Superiority or Other; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-19.4 to 16.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Group 3: Belatacept Less Intensive (LI) + MMF vs Group 5: Tacrolimus; Analysis at Month 12; Test type: Superiority or Other; Mean Difference (Final Values) = -10.8, 95% CI 2-sided [-29.3 to 7.9] — [estimate comment as in outcome 1, analysis 1]

45. Primary Outcome: Number of Participants Who Had Adverse Events (AEs), Death, Serious AEs (SAEs) or Were Discontinued Due to AEs (Includes Long Term Extension [LTE] Data)
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition in a subject administered an investigational product and that does not necessarily have a causal relationship with this treatment. SAE=any untoward medical occurrence that results in death, is life-threatening, requires or prolongs inpatient hospitalization (including elective surgery), results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an important medical event.
Time Frame: Day 1 (randomization) to Week 104 + within 56 Days after the last infusion/dose, Deaths were monitored up to database lock (20-June-2011)
Population: ITT-LTE population, (all randomized and transplanted participants who entered long term extension). Participants were grouped according to the treatment to which they were randomized initially.
Measure: Number; unit: participants
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 30 | 27 | 24 | 38 | 26
participants
  SAEs | 18 | 22 | 17 | 29 | 21
  Related SAEs | 5 | 9 | 9 | 12 | 9
  Discontinued due to SAEs | 2 | 4 | 1 | 1 | 0
  AEs | 30 | 27 | 23 | 38 | 26
  Related AEs | 27 | 21 | 20 | 33 | 23
  Discontinued due to AEs | 2 | 5 | 1 | 1 | 0
  Deaths (due to AE) | 2 | 3 | 1 | 3 | 0
  Deaths (not due to AE) | 0 | 1 | 0 | 0 | 0

46. Primary Outcome: Number of Participants Who Had AEs of Special Interest During the LTE
Description: AE of special interest included malignancies (including skin carcinomas), infections (viral, cytomegalovirus, herpes, fungal, and bacterial).
Time Frame: Day 1 (randomization) through database lock (20-June-2011)
Population: ITT-LTE population, all randomized and transplanted participants who entered long term extension
Measure: Number; unit: participants
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 30 | 27 | 24 | 38 | 26
participants
  Malignancies | 1 | 4 | 3 | 8 | 3
  Infections and Infestations | 8 | 6 | 9 | 11 | 8

47. Primary Outcome: Number of Participants With Marked Hematology Abnormalities During the LTE
Description: Low platelet count: <50*10^9 c/µl; Low leukocytes: <2.0*10^3 c/µl; Low lymphocytes (absolute): <0.5*10^3 c/µl; Low neutrophils (absolute): <1.0*10^3 c/µl.
Time Frame: Every 4 weeks from Week 53 to Week 104.
Population: ITT-LTE population: All randomized and transplanted participants who entered long-term extension. n= participants who had a laboratory test reading after transplant for the specific analyte.
Measure: Number; unit: participants
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 30 | 27 | 24 | 38 | 26
participants
  Low Platelets: (n=29, 26, 22, 37, 25) | 1 | 2 | 0 | 2 | 0
  Low Leukocytes : (n=29, 27, 22, 37, 25) | 1 | 2 | 0 | 3 | 0
  Low Absolute Lymphocyte: (n=29, 27, 22, 36, 25) | 8 | 3 | 3 | 5 | 3
  Low Absolute Neutrophils: (n=29, 27, 22, 36, 25) | 0 | 2 | 1 | 2 | 0

48. Primary Outcome: Number of Participants With Marked Liver and Kidney Function Abnormalities During the LTE
Description: ULN= upper limit of normal; Normal ranges are provided by the Central Laboratory and may vary according to sex and age. High alanine aminotransferase (ALT): >5.0*ULN U/L; High aspartate aminotransferase (AST): >5.0*ULN U/L; High direct bilirubin: >3.0*ULN mg/dL; High g-glutamyl transferase (GGT): >5.0*ULN U/L; High total bilirubin: >3.0*ULN mg/dL; High creatinine: > 3.0*ULN mg/dL
Time Frame: Every 4 weeks from Week 53 to Week 104.
Population: as for outcome 47
Measure: Number; unit: participants
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 29 | 27 | 22 | 37 | 25
participants
  High ALT | 0 | 2 | 1 | 4 | 3
  High AST | 0 | 3 | 2 | 4 | 3
  High Direct Bilirubin | 1 | 4 | 1 | 3 | 2
  High GGT | 2 | 6 | 6 | 13 | 8
  High Total Bilirubin | 1 | 3 | 1 | 2 | 0
  High Creatinine | 0 | 0 | 0 | 1 | 0

49. Primary Outcome: Number of Participants With Marked Electrolytes, Protein and Metabolic Test Abnormalities During the LTE
Description: Low Serum Potassium: <3.0 meq/L; High serum potassium:>6.0 mEq/L; Low serum magnesium:<0.8 mEq/L; Low serum sodium: <130 mEq/L; High serum sodium: >155 mEq/L; Low inorganic phosphorus: <2.0 mg/dL; High uric acid: >10 mg/dL
Time Frame: Every 4 weeks from Week 53 to Week 104.
Population: as for outcome 47
Measure: Number; unit: participants
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 29 | 27 | 22 | 37 | 25
participants
  Low Serum Potassium | 0 | 0 | 0 | 0 | 0
  High Serum Potassium | 1 | 1 | 0 | 0 | 0
  Low Serum Sodium | 1 | 2 | 1 | 1 | 0
  High Serum Sodium | 0 | 0 | 1 | 0 | 0
  Low Inorganic Phosphorus | 1 | 0 | 1 | 1 | 0
  High Uric Acid | 0 | 1 | 0 | 6 | 6

50. Secondary Outcome: Number of Participants Who Received Anti-hypertensive Therapy at Month 12
Time Frame: 12 months posttransplant
Population: ITT population, all randomized and transplanted participants.
Measure: Number; unit: participants
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept Less Intensive (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 41 | 39 | 36 | 48 | 42
participants
  Received at least 1 medication | 20 | 19 | 14 | 26 | 21
  Received 1 medication | 13 | 16 | 8 | 17 | 12
  Received 2 medications | 6 | 2 | 2 | 5 | 5
  Received 3 medications | 1 | 1 | 4 | 3 | 3
  Received 4 medications | 1 | 0 | 0 | 1 | 1

51. Secondary Outcome: Percentage of Participants With New Onset Diabetes Mellitus (NODM): 12-month Treatment Phase
Description: A participant who did not have diabetes prior to randomization was determined to have NODM if(i) the participant received an antidiabetic medication for a duration of at least 30 days or(ii) at least two fasting plasma glucose (FPG) tests indicate that FPG is>=126 mg/dL (7.0 mmol/L). For 95% CI within each group, normal approximation is used if N>=5. For 95% CI of difference, adjustment is made for randomization strata (HCV-Infection status at baseline) if N >= 5 in each treatment arm.
Time Frame: 6 and 12 months posttransplant
Population: ITT population, all randomized participants without Diabetes Mellitus (pre-transplantation).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 31 | 32 | 36 | 38 | 37
percentage of participants
  6 months | 35.5 [18.6 to 52.3] | 15.6 [3.0 to 28.2] | 13.9 [2.6 to 25.2] | 21.1 [8.1 to 34.0] | 35.1 [19.8 to 50.5]
  12 months | 35.5 [18.6 to 52.3] | 15.6 [3.0 to 28.2] | 13.9 [2.6 to 25.2] | 23.7 [10.2 to 37.2] | 37.8 [22.2 to 53.5]
Statistical Analysis 1: Comparison: Group 1: Basiliximab+Belatacept (MI) + MMF vs Group 4: Tacrolimus + MMF; Analysis at Month 6; Test type: Superiority or Other; Mean Difference (Final Values) = 14.4, 95% CI 2-sided [-6.3 to 36.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Group 2: Belatacept (MI) + MMF vs Group 4: Tacrolimus + MMF; Analysis at Month 6; Test type: Superiority or Other; Mean Difference (Final Values) = -5.4, 95% CI 2-sided [-23.4 to 10.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Group 3: Belatacept (LI) + MMF vs Group 4: Tacrolimus + MMF; Analysis at Month 6; Test type: Superiority or Other; Mean Difference (Final Values) = -7.2, 95% CI 2-sided [-23.4 to 10.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Group 1: Basiliximab+Belatacept (MI) + MMF vs Group 5: Tacrolimus; Analysis at Month 6; Test type: Superiority or Other; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-22.0 to 23.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Group 2: Belatacept (MI) + MMF vs Group 5: Tacrolimus; Analysis at Month 6; Test type: Superiority or Other; Mean Difference (Final Values) = -19.5, 95% CI 2-sided [-38.6 to -0.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Group 3: Belatacept (LI) + MMF vs Group 5: Tacrolimus; Analysis at Month 6; Test type: Superiority or Other; Mean Difference (Final Values) = -21.2, 95% CI 2-sided [-39.1 to -1.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Group 1: Basiliximab+Belatacept (MI) + MMF vs Group 4: Tacrolimus + MMF; Analysis at Month 12; Test type: Superiority or Other; Mean Difference (Final Values) = 11.8, 95% CI 2-sided [-8.7 to 34.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Group 2: Belatacept (MI) + MMF vs Group 5: Tacrolimus; Analysis at Month 12; Test type: Superiority or Other; Mean Difference (Final Values) = -8.1, 95% CI 2-sided [-25.2 to 8.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Group 3: Belatacept (LI) + MMF vs Group 4: Tacrolimus + MMF; Analysis at Month 12; Test type: Superiority or Other; Mean Difference (Final Values) = -9.8, 95% CI 2-sided [-26.3 to 7.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Group 1: Basiliximab+Belatacept (MI) + MMF vs Group 5: Tacrolimus; Analysis at Month 12; Test type: Superiority or Other; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-24.5 to 21.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Group 2: Belatacept (MI) + MMF vs Group 5: Tacrolimus; Analysis at Month 12; Test type: Superiority or Other; Mean Difference (Final Values) = -22.2, 95% CI 2-sided [-40.5 to -1.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Group 3: Belatacept (LI) + MMF vs Group 5: Tacrolimus; Analysis at Month 12; Test type: Superiority or Other; Mean Difference (Final Values) = -23.9, 95% CI 2-sided [-41.8 to -4.3] — [estimate comment as in outcome 1, analysis 1]

52. Secondary Outcome: Glycosylated Hemoglobin (HbA1C) Values: 12-month Treatment Phase
Description: The HbA1c test is important in diabetes as a long-term measure of control over blood glucose, where the glucose bound to hemoglobin during the past 3-4 months is measured. A baseline diabetes participant was one who had a medical history of diabetes or being under anti-diabetic medication at the time of the transplantation. BL = baseline, DM = Diabetes mellitus.
Time Frame: 6, 12 months (mth) posttransplant
Population: ITT population, all randomized and transplanted participants. n = Participants with both baseline and postbaseline values.
Measure: Mean (Standard Deviation); unit: Percentage of glycosylated hemoglobin
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept Less Intensive (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 50 | 48 | 49 | 53 | 50
Percentage of glycosylated hemoglobin
  6 mo: All participants (n=39, 34, 38, 47, 35) | 5.8 (1.07) | 5.8 (0.96) | 5.6 (0.75) | 5.4 (0.90) | 5.4 (0.84)
  6 mo: DM at BL (n=15, 12, 10, 12, 10) | 6.5 (1.19) | 6.6 (1.02) | 6.1 (0.76) | 5.8 (1.19) | 5.4 (0.59)
  6 mo: DM at BL/DM at 6m (n=23, 14, 14, 19, 18) | 6.1 (1.17) | 6.4 (1.02) | 5.9 (0.90) | 5.5 (1.04) | 5.4 (0.62)
  12 mo: All participants (n=40, 35, 35, 44, 37) | 6.0 (1.32) | 5.8 (1.03) | 5.7 (0.97) | 5.5 (0.76) | 5.8 (1.85)
  12 mo: DM at BL (n=15, 11, 7, 11, 12) | 6.9 (1.60) | 6.7 (1.40) | 6.7 (1.49) | 6.2 (0.96) | 6.5 (3.05)
  12 mo: DM at BL/DM at 12 mth (n=23,13 ,11,18,20) | 6.3 (1.58) | 6.6 (1.29) | 6.2 (1.40) | 6.0 (0.84) | 6.3 (2.39)

53. Secondary Outcome: Number of Participants Who Had AEs, Death, SAEs or Were Discontinued Due to AEs: 12-month Treatment Phase
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition in a participant administered an investigational product and that does not necessarily have a causal relationship with this treatment. SAE=any untoward medical occurrence that results in death, is life-threatening, requires or prolongs inpatient hospitalization (including elective surgery), results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an important medical event
Time Frame: Day 1 (randomization) to 12 m + 8 week follow-up or ≤ 56 days after discontinuation of study medication
Population: ITT population: all randomized and transplanted participants
Measure: Number; unit: participants
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 50 | 48 | 49 | 53 | 50
participants
  Death | 4 | 4 | 9 | 1 | 4
  SAEs | 28 | 29 | 37 | 40 | 35
  Related SAEs | 12 | 11 | 14 | 16 | 19
  Discontinued due to SAEs | 7 | 6 | 11 | 4 | 13
  AEs | 50 | 48 | 48 | 53 | 50
  Related AEs | 45 | 34 | 33 | 42 | 42
  Discontinued due to AEs | 7 | 7 | 12 | 7 | 18

54. Secondary Outcome: Number of Participants Who Had Adverse Events of Special Interest During 12-month Treatment Phase
Description: AE of of special interest included malignancies (including skin carcinomas), infections (viral, cytomegalovirus, herpes, fungal, and bacterial), serious infections
Time Frame: Day 1 (randomization) to 12 months or ≤ 56 days after discontinuation of study medication
Population: ITT population, all randomized and transplanted participants.
Measure: Number; unit: participants
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 50 | 48 | 49 | 53 | 50
participants
  Malignancies | 1 | 0 | 2 | 2 | 2
  Post-transplant lymphoproliferative disorder | 0 | 0 | 1 | 0 | 0
  All Infections | 32 | 39 | 30 | 31 | 29
  Bacterial infections | 5 | 11 | 11 | 6 | 13
  Fungal infections | 6 | 9 | 14 | 6 | 5
  Viral infections | 10 | 11 | 14 | 9 | 7
  Cytomegalovirus infections | 5 | 4 | 10 | 4 | 1
  Polyoma virus infections | 0 | 1 | 0 | 0 | 0
  Herpes infections | 3 | 3 | 4 | 3 | 2
  Hepatitis C virus recurrence | 14 | 7 | 6 | 13 | 9
  Serious infections | 11 | 12 | 13 | 12 | 12
  Autoimmune events | 0 | 0 | 1 | 0 | 2
  Acute peri-infusional events | 5 | 1 | 0 | NA | NA
  Thrombotic and embolic events | 3 | 3 | 7 | 10 | 5

55. Secondary Outcome: Number of Participants With Marked Hematology Abnormalities: 12-month Treatment Phase
Description: Low hemoglobin: <8 g/dL; Low platelet count: <50*10^9 C/L; Low leukocytes: <2.0 *10^3 c/µL; Low lymphocytes (absolute): <0.5*10^3 c/µL; Low neutrophils (absolute): <1.0*10^3 Cc/µL.
Time Frame: Baseline (pretransplant), 2, 4, 8, 12 weeks, and every 4 weeks for week 16 to 52
Population: ITT population, all randomized and transplanted participants. n= participants with all observations.
Measure: Number; unit: participants
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 50 | 48 | 49 | 53 | 50
participants
  Low Hemoglobin: (n=48, 46, 44, 52, 50) | 2 | 6 | 2 | 0 | 6
  Low Platelets: (n=48, 46, 43, 52, 50) | 0 | 1 | 4 | 2 | 2
  Low Leukocytes : (n=48, 46, 44, 52, 50) | 6 | 6 | 5 | 4 | 3
  Low Absolute Lymphocyte: (n=48, 46, 44, 52, 50) | 29 | 18 | 26 | 17 | 16
  Low Absolute Neutrophils : (n=48, 46, 44, 52, 50) | 6 | 4 | 4 | 8 | 1

56. Secondary Outcome: Number of Participants With Marked Liver and Kidney Function Abnormalities: 12-month Treatment Phase
Description: ULN= upper limit of normal; Normal ranges are provided by the central laboratory and may vary according to sex and age. High alkaline phosphatase (ALP): >5.0*ULN U/L; High alanine aminotransferase (ALT): >5.0*ULN U/L; High aspartate aminotransferase (AST): >5.0*ULN U/L; High direct bilirubin: >3.0 * ULN mg/dL; High g-glutamyl transferase (GGT): >5.0*ULN U/L; High total bilirubin: >3.0*ULN mg/dL; High creatinine: > 3.0*ULN mg/dL
Time Frame: Baseline (pretransplant), 4, 12, 24, 52 weeks
Population: ITT population, all randomized and transplanted participants. n= participants with all observations.
Measure: Number; unit: participants
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 50 | 48 | 49 | 53 | 50
participants
  High ALP: (n=48, 47, 44, 53, 50) | 5 | 6 | 6 | 4 | 6
  High ALT: (n=48, 47, 44, 53, 50) | 16 | 18 | 19 | 16 | 9
  High AST: (n=48, 47, 44, 53, 50) | 9 | 14 | 16 | 8 | 2
  High Direct Bilirubin: (n=48, 47, 44, 53, 50) | 15 | 18 | 19 | 20 | 16
  High GGT: (n=48, 47, 44, 53, 50) | 25 | 24 | 24 | 27 | 22
  High Total Bilirubin: (n=48, 47, 44, 53, 50) | 9 | 13 | 16 | 12 | 10
  High Creatinine: (n=47, 44, 44, 53, 50) | 0 | 0 | 0 | 0 | 0

57. Secondary Outcome: Number of Participants With Marked Electrolytes, Protein and Metabolic Test Abnormalities: 12-month Treatment Phase
Description: Low total calcium: <7 mg/dL; High total calcium: >12.5 mg/dL ; Low bicarbonate: <11 mEq/L; Low serum potassium: <3.0 mEq/L; High serum potassium:>6.0 mEq/L; High serum magnesium: >2.46 mEq/L; Low serum magnesium:<0.8 mEq/L; Low serum sodium: <130 mEq/L; High serum sodium: >155 mEq/L; Low inorganic phosphorus: <2.0 mg/dL; Low albumin: <2 g/dL; High uric acid: >10 mg/dL
Time Frame: Baseline (pretransplant), Weeks 4, 12, 24, and 52
Population: ITT population, all randomized and transplanted participants. n= participants with all observations.
Measure: Number; unit: participants
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 50 | 48 | 49 | 53 | 50
participants
  Low Total Calcium (n=48, 47, 44, 53, 50) | 0 | 1 | 1 | 1 | 0
  High Total Calcium (n=48, 47, 44, 53, 50) | 0 | 0 | 0 | 0 | 0
  Low Bicarbonate (n=47, 47, 44, 53, 50) | 0 | 0 | 0 | 1 | 0
  Low Serum Potassium (n=48, 47, 44, 53, 50) | 0 | 2 | 1 | 1 | 0
  High Serum Potassium (n=48, 47, 44, 53, 50) | 1 | 0 | 1 | 2 | 1
  High Serum Magnesium (n=48, 47, 44, 53, 50) | 0 | 0 | 0 | 0 | 0
  Low Serum Magnesium (n=48, 47, 44, 53, 50) | 2 | 0 | 2 | 0 | 1
  Low Serum Sodium (n=48, 47, 44, 53, 50) | 3 | 2 | 2 | 2 | 2
  High Serum Sodium (n=48, 47, 44, 53, 50) | 0 | 0 | 0 | 0 | 0
  Low Inorganic Phosphorus (n=48, 47, 44, 53, 50) | 0 | 2 | 1 | 2 | 0
  Low Albumin (n=47, 47, 45, 53, 50) | 2 | 1 | 0 | 0 | 0
  High Uric Acid (n=48, 47, 44, 53, 50) | 2 | 1 | 2 | 5 | 5

58. Secondary Outcome: Number of Participants Who Had Abnormalities in Electrocardiograms: 12-month Treatment Phase
Time Frame: Baseline (pretransplant), Week 52
Population: ECG data was not analyzed.
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

59. Secondary Outcome: Change in Protein to Creatinine Ratio From Month 3 to Month 12.
Time Frame: Month 3 and 12
Population: Protein creatinine ratio change was not analyzed
Arm/Group | Group 1: Basiliximab+Belatacept (MI) + MMF | Group 2: Belatacept (MI) + MMF | Group 3: Belatacept (LI) + MMF | Group 4: Tacrolimus + MMF | Group 5: Tacrolimus
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Basiliximab+Belatacept (MI)+Mycophenolate Mofetil (MMF) | MI+MMF | Belaticept (LI) + MMF | Tacrolimus | Tacrolimus + MMF
Serious Adverse Events (participants affected / at risk) | 18/30 | 17/24 | 22/27 | 21/26 | 29/38
Other Adverse Events (participants affected / at risk) | 29/30 | 23/24 | 27/27 | 25/26 | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Basiliximab+Belatacept (MI)+Mycophenolate Mofetil (MMF) (N=30) | MI+MMF (N=24) | Belaticept (LI) + MMF (N=27) | Tacrolimus (N=26) | Tacrolimus + MMF (N=38)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 2 | 2
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 1 | 1
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Coeliac artery stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 2
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Intra-abdominal haemorrhage (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Liver abscess (Infections and infestations) | 1 | 1 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 1 | 2
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 5 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Arterial thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Biliary ischaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Biloma (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Device leakage (General disorders) | 0 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Epstein-Barr virus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Haematocrit decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0 | 3
Medical device complication (General disorders) | 0 | 0 | 0 | 1 | 0
Parvovirus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Retinal vein occlusion (Eye disorders) | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0 | 0 | 1
Status epilepticus (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Tracheobronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2
Alcoholism (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Artery dissection (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1
Biliary abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1
Encephalomalacia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 1 | 2 | 4 | 3
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Volvulus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 3 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Arterial insufficiency (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 1 | 1 | 2 | 0 | 2
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Epididymitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 1
Hepatic artery thrombosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 1
Hepatopulmonary syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Hernia (General disorders) | 1 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 2 | 4
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Bile duct stenosis (Hepatobiliary disorders) | 3 | 3 | 0 | 2 | 2
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 1
Cholangitis (Hepatobiliary disorders) | 2 | 2 | 1 | 2 | 5
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Haemobilia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Hepatic neoplasm malignant recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2
Hepatitis B (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Hepatitis C (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 2 | 1 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Cytomegalovirus viraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Gynaecomastia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Hepatic artery stenosis (Hepatobiliary disorders) | 1 | 0 | 1 | 2 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Hepatic haemorrhage (Hepatobiliary disorders) | 0 | 2 | 0 | 0 | 0
Incision site cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Meningitis aseptic (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Mental disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Nephropathy toxic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0
Pleura carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 1 | 0 | 0
Transplant rejection (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 2 | 0 | 0 | 0
Varicella (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 1 | 0
Biliary anastomosis complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Groin abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Hepatic haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 3 | 2 | 0 | 0 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1
Transient psychosis (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Biliary tract disorder (Hepatobiliary disorders) | 1 | 0 | 1 | 1 | 0
Body temperature increased (Investigations) | 1 | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 1 | 0
Convulsion (Nervous system disorders) | 1 | 1 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 2
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Drug dispensing error (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Epstein-Barr virus associated lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 0 | 0
Hepatitis E (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Multi-organ failure (General disorders) | 1 | 0 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Portal vein stenosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 2 | 1 | 1 | 1
Salivary gland fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Basiliximab+Belatacept (MI)+Mycophenolate Mofetil (MMF) (N=30) | MI+MMF (N=24) | Belaticept (LI) + MMF (N=27) | Tacrolimus (N=26) | Tacrolimus + MMF (N=38)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 13 | 5 | 11 | 11 | 14
Ascites (Gastrointestinal disorders) | 9 | 4 | 6 | 5 | 9
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 3 | 2 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 1 | 2 | 0 | 0
Bloody discharge (General disorders) | 2 | 0 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 0 | 2 | 0 | 0
Fatigue (General disorders) | 11 | 2 | 4 | 12 | 12
Fungal skin infection (Infections and infestations) | 2 | 1 | 3 | 0 | 0
Gait disturbance (General disorders) | 1 | 2 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 2 | 2 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 1 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 3 | 2 | 3 | 4 | 2
Incision site erythema (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 7 | 5 | 8 | 9 | 8
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0 | 0
Intra-abdominal haemorrhage (Vascular disorders) | 0 | 0 | 1 | 2 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2
Mental status changes (Psychiatric disorders) | 1 | 0 | 2 | 2 | 0
Nasopharyngitis (Infections and infestations) | 6 | 3 | 9 | 2 | 10
Nausea (Gastrointestinal disorders) | 8 | 7 | 8 | 9 | 13
Oedema (General disorders) | 2 | 5 | 3 | 0 | 3
Osteopenia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 1 | 3
Platelet count decreased (Investigations) | 2 | 1 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 2 | 0 | 1 | 3 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 2
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 0
Visual acuity reduced (Eye disorders) | 3 | 1 | 1 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 2 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 5 | 4 | 8 | 6
Blood glucose increased (Investigations) | 2 | 0 | 0 | 0 | 5
Bronchitis (Infections and infestations) | 0 | 2 | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 12 | 7 | 10 | 10 | 14
Decreased appetite (Metabolism and nutrition disorders) | 4 | 4 | 3 | 6 | 6
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 3 | 2 | 2 | 2
Dysuria (Renal and urinary disorders) | 0 | 2 | 4 | 1 | 2
Facial paresis (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 2 | 1 | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 2 | 1 | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 4 | 2 | 2 | 1 | 4
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 1 | 0 | 2
Nocturia (Renal and urinary disorders) | 1 | 1 | 2 | 2 | 1
Oral herpes (Infections and infestations) | 2 | 1 | 2 | 0 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 5 | 2 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 5 | 5 | 7 | 6
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2 | 0 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
Tremor (Nervous system disorders) | 1 | 3 | 2 | 10 | 14
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 3
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 1 | 0 | 2
Abdominal hernia (Gastrointestinal disorders) | 2 | 0 | 2 | 0 | 3
Bacteraemia (Infections and infestations) | 2 | 0 | 0 | 1 | 2
Blood pressure increased (Investigations) | 2 | 1 | 0 | 1 | 1
Cataract (Eye disorders) | 2 | 1 | 0 | 1 | 2
Clostridial infection (Infections and infestations) | 0 | 0 | 2 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 2 | 8 | 3 | 6
Dyspepsia (Gastrointestinal disorders) | 2 | 1 | 3 | 3 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 6 | 7 | 5
Enterococcal infection (Infections and infestations) | 0 | 0 | 3 | 0 | 3
Gamma-glutamyltransferase increased (Investigations) | 1 | 2 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 1 | 2 | 1 | 3
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 3 | 3 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1 | 4 | 1 | 1
Hyporeflexia (Nervous system disorders) | 0 | 0 | 0 | 1 | 2
Irritability (General disorders) | 1 | 0 | 0 | 3 | 2
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1 | 3
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Lymphocele (Vascular disorders) | 2 | 0 | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 2
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0 | 3
Procedural pain (Injury, poisoning and procedural complications) | 10 | 5 | 9 | 9 | 12
Proteinuria (Renal and urinary disorders) | 4 | 1 | 1 | 4 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3 | 3 | 2
Renal failure acute (Renal and urinary disorders) | 2 | 0 | 2 | 2 | 8
Rib fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 1 | 1 | 2
Urine output decreased (Investigations) | 2 | 0 | 1 | 4 | 2
White blood cell count increased (Investigations) | 0 | 0 | 3 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 10 | 3 | 8 | 9 | 13
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 1 | 2 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 7 | 9 | 6 | 11
Bacterial test positive (Investigations) | 0 | 0 | 0 | 1 | 3
Blood potassium increased (Investigations) | 0 | 0 | 0 | 3 | 1
Bradycardia (Cardiac disorders) | 0 | 1 | 2 | 5 | 2
Candidiasis (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 3 | 2 | 0 | 5
Cytomegalovirus infection (Infections and infestations) | 2 | 3 | 2 | 0 | 3
Dizziness (Nervous system disorders) | 6 | 1 | 4 | 3 | 4
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 1 | 3
Eye pruritus (Eye disorders) | 0 | 0 | 2 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 1 | 1 | 2
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 12 | 4 | 9 | 14 | 10
Herpes zoster (Infections and infestations) | 0 | 3 | 2 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 2 | 3 | 8 | 8
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 1 | 2 | 0 | 0
Hypotension (Vascular disorders) | 5 | 1 | 7 | 6 | 7
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 1 | 1
Incision site complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2
Influenza (Infections and infestations) | 1 | 0 | 2 | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 2 | 3 | 2
Liver function test abnormal (Investigations) | 6 | 1 | 3 | 9 | 7
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 2
Mood swings (Psychiatric disorders) | 1 | 1 | 0 | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 3 | 3 | 2 | 7
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 4 | 3
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 1 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 1 | 3 | 8 | 10
Renal tubular necrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 2
Seasonal allergy (Immune system disorders) | 0 | 1 | 0 | 2 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0
Staphylococcus test positive (Investigations) | 1 | 0 | 0 | 2 | 1
Toothache (Gastrointestinal disorders) | 2 | 1 | 1 | 2 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 3 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 4
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 1
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 3
Bile duct stenosis (Hepatobiliary disorders) | 3 | 0 | 2 | 4 | 1
Breath sounds abnormal (Investigations) | 3 | 2 | 3 | 3 | 3
C-reactive protein increased (Investigations) | 0 | 1 | 2 | 1 | 1
Catheter site pain (General disorders) | 0 | 1 | 2 | 0 | 0
Chest pain (General disorders) | 2 | 4 | 4 | 2 | 1
Chills (General disorders) | 3 | 0 | 3 | 1 | 3
Cholangitis (Hepatobiliary disorders) | 1 | 1 | 1 | 0 | 4
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 4 | 2 | 3 | 9
Diarrhoea (Gastrointestinal disorders) | 12 | 10 | 10 | 11 | 23
Excoriation (Injury, poisoning and procedural complications) | 1 | 1 | 3 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 3 | 0
Flatulence (Gastrointestinal disorders) | 4 | 2 | 1 | 2 | 2
Flushing (Vascular disorders) | 0 | 0 | 1 | 0 | 2
Generalised oedema (General disorders) | 1 | 1 | 3 | 3 | 2
Haematuria (Renal and urinary disorders) | 2 | 1 | 1 | 1 | 1
Hepatitis C (Infections and infestations) | 2 | 2 | 0 | 1 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 1 | 4 | 6 | 8
Impaired healing (General disorders) | 1 | 1 | 2 | 2 | 0
Laryngitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 1 | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 4 | 0 | 3
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 3
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 2 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 2 | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 5 | 2 | 4 | 5 | 5
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1 | 5 | 2
Respiratory tract infection (Infections and infestations) | 2 | 0 | 1 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 1 | 2 | 1 | 3
Varices oesophageal (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Vision blurred (Eye disorders) | 3 | 0 | 2 | 1 | 1
Visual impairment (Eye disorders) | 2 | 0 | 2 | 0 | 2
Weight increased (Investigations) | 5 | 6 | 2 | 6 | 3
White blood cell count decreased (Investigations) | 3 | 1 | 1 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 3 | 3 | 3 | 4 | 4
Agitation (Psychiatric disorders) | 2 | 0 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 1 | 0 | 0
Asthenia (General disorders) | 4 | 3 | 4 | 3 | 2
Blood bilirubin increased (Investigations) | 4 | 0 | 1 | 0 | 2
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 2 | 0 | 1
Cholestasis (Hepatobiliary disorders) | 2 | 0 | 2 | 3 | 6
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 3
Ear infection (Infections and infestations) | 0 | 2 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 3 | 3 | 1 | 0
Enterococcus test positive (Investigations) | 0 | 0 | 1 | 2 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 2 | 2 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 1 | 3 | 2
Gastritis (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 2
Hallucination (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0
Hepatic artery stenosis (Hepatobiliary disorders) | 1 | 1 | 2 | 1 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 | 1 | 1 | 2
Hypertension (Vascular disorders) | 5 | 6 | 6 | 11 | 16
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 0
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1 | 0
Influenza like illness (General disorders) | 1 | 1 | 1 | 3 | 2
Leukopenia (Blood and lymphatic system disorders) | 8 | 9 | 5 | 3 | 13
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 3 | 1 | 3 | 2 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 2 | 0 | 0
Oedema peripheral (General disorders) | 11 | 7 | 10 | 10 | 19
Pain (General disorders) | 4 | 2 | 1 | 1 | 4
Paraesthesia (Nervous system disorders) | 3 | 0 | 1 | 2 | 3
Periodontitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 | 5 | 6 | 8 | 10
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 3 | 0 | 1
Transaminases increased (Investigations) | 3 | 1 | 3 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 2 | 4 | 0 | 2
Urinary tract infection (Infections and infestations) | 7 | 4 | 8 | 2 | 5
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 1 | 0 | 3
Abdominal distension (Gastrointestinal disorders) | 7 | 3 | 3 | 2 | 5
Alanine aminotransferase increased (Investigations) | 0 | 2 | 1 | 1 | 1
Anastomotic stenosis (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0
Biliary anastomosis complication (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 3 | 1 | 2 | 0 | 0
Blood triglycerides increased (Investigations) | 2 | 2 | 0 | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 1 | 1 | 2 | 1 | 0
Confusional state (Psychiatric disorders) | 3 | 0 | 1 | 2 | 0
Device related infection (Infections and infestations) | 1 | 0 | 1 | 3 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 2 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 1 | 2 | 0 | 1
Hepatic haematoma (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 1 | 2
Hot flush (Vascular disorders) | 4 | 1 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 11 | 5 | 9 | 5 | 9
Incision site pain (Injury, poisoning and procedural complications) | 5 | 2 | 2 | 4 | 6
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1
Malaise (General disorders) | 0 | 0 | 1 | 2 | 4
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2 | 2 | 2
Nephrolithiasis (Renal and urinary disorders) | 2 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 4 | 3 | 1 | 3
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 2 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 1 | 1
Pharyngitis (Infections and infestations) | 0 | 2 | 1 | 0 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 1 | 2 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 2 | 5 | 5
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 3 | 2 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Transient psychosis (Psychiatric disorders) | 0 | 0 | 0 | 1 | 2
Urinary incontinence (Renal and urinary disorders) | 1 | 1 | 0 | 2 | 1
Wound complication (Injury, poisoning and procedural complications) | 3 | 0 | 1 | 1 | 3
Wound infection (Infections and infestations) | 4 | 1 | 3 | 2 | 0
Wound secretion (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1 | 0
Amnesia (Nervous system disorders) | 2 | 0 | 0 | 2 | 2
Anxiety (Psychiatric disorders) | 7 | 1 | 3 | 6 | 7
Blood creatinine increased (Investigations) | 5 | 1 | 2 | 6 | 8
Blood magnesium decreased (Investigations) | 1 | 0 | 0 | 0 | 2
Body temperature increased (Investigations) | 2 | 0 | 1 | 0 | 0
Clostridium test positive (Investigations) | 0 | 0 | 2 | 0 | 2
Convulsion (Nervous system disorders) | 0 | 1 | 1 | 1 | 2
Cystitis (Infections and infestations) | 0 | 2 | 0 | 0 | 1
Depression (Psychiatric disorders) | 10 | 4 | 2 | 6 | 5
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 4 | 3
Hepatic enzyme increased (Investigations) | 5 | 4 | 4 | 1 | 4
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 0 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 0 | 4 | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 9 | 8 | 3 | 8
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2
Incision site haemorrhage (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 1 | 1
Jaundice (Hepatobiliary disorders) | 0 | 2 | 1 | 2 | 2
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 0 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 1 | 3 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0 | 1
Oliguria (Renal and urinary disorders) | 2 | 1 | 1 | 4 | 1
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 2
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1 | 0 | 2 | 0
Post procedural discharge (Injury, poisoning and procedural complications) | 2 | 0 | 3 | 0 | 2
Pyrexia (General disorders) | 11 | 8 | 10 | 8 | 9
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2 | 1
Scrotal oedema (Reproductive system and breast disorders) | 2 | 2 | 0 | 1 | 2
Sleep disorder (Psychiatric disorders) | 0 | 1 | 2 | 3 | 2
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 4 | 0 | 4 | 2 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 6 | 3 | 1 | 6
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2 | 0
Vomiting (Gastrointestinal disorders) | 6 | 4 | 4 | 8 | 10
Weight decreased (Investigations) | 3 | 3 | 1 | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.